CLINICAL TRIAL: NCT03502616
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, STUDY OF THE EFFICACY AND SAFETY OF TOFACITINIB IN SUBJECTS WITH ACTIVE ANKYLOSING SPONDYLITIS (AS)
Brief Title: Efficacy and Safety of Tofacitinib in Subjects With Active Ankylosing Spondylitis (AS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921120; AS (Other: Alias Study Number); 2018-000226-58 (EudraCT Number)
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tofacitinib (Experimental)
  Interventions: Drug: Tofacitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Oral administration twice per day

SUMMARY:
The purpose of this study is to determine if tofacitinib is safe and effective in subjects with active ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Ankylosing Spondylitis (AS) based on the Modified New York Criteria for AS (1984).
* Must have a radiograph of SI joints (AP Pelvis) documenting diagnosis of AS.
* Has active disease despite nonsteroidal anti-inflammatory drug (NSAID) therapy or intolerant to NSAIDs.

Exclusion Criteria:

* History of known or suspected complete ankylosis of the spine.
* History of allergies, intolerance or hypersensitivity to lactose or tofacitinib.
* History of any other rheumatic disease.
* Any subject with condition affecting oral drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (99):
- United States (28):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Gilbert, Arizona
  - Medvin Clinical Research, Covina, California
  - Rheumatology Center of San Diego PC, San Diego, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Robin K. Dore, MD, Inc., Tustin, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Advanced Radiology, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Southcoast Research Center, Inc., Miami, Florida
  - Millennium Research, Ormond Beach, Florida
  - Bluegrass Community Research, Inc, Lexington, Kentucky
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - M3-Emerging Medical Research, LLC, Durham, North Carolina
  - Paramount Medical Research and Consulting, LLC, Middleburg Heights, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology, Summerville, South Carolina
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Adriana Pop-Moody MD - Clinic PA, Corpus Christi, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Clinical Research Unit, Houston, Texas
  - Investigational Drug Services, Houston, Texas
  - Memorial Hermann Hospital Imaging, Houston, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Trinity Universal Research Associates, Inc., Plano, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Australia (7):
  - Pacific Radiology,, Maroochydore, Queensland
  - Rheumatology Research Unit Sunshine Coast, Maroochydore, Queensland
  - Emeritus Research Pty. Ltd., Camberwell, Victoria
  - Melbourne Radiology Clinic, East Melbourne, Victoria
  - SKG Radiology, Subiaco, Western Australia
  - Western Cardiology, Subiaco, Western Australia
  - RK Will Pty Ltd, Victoria Park, Western Australia
- Bulgaria (3):
  - Multiprofile Hospital for active treatment "Kaspela" EOOD, Plovdiv
  - Diagnostic-Consulting Center XVII - Sofia, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
- Canada (2):
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- China (5):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hosptial of Wenzhou Medical University, Wenzhou, Zhejiang
  - Rheumatology and Immunology Department, Shanghai Changzheng Hospital, Shanghai
- Czechia (7):
  - Lekarna Rezidence Nova Karolina, Ostrava
  - CCBR Ostrava s.r.o., Ostrava
  - BENU Lekarna, Pardubice
  - CCR, Czech a.s., Pardubice
  - Lekarna Hradebni, s.r.o., Uherské Hradiště
  - Uherskohradistska nemocnice, a.s., Uherské Hradiště
  - Medical Plus s.r.o., Uherské Hradiště
- CHRU de Tours, Hopital Trousseau, Tours, France
- Hungary (3):
  - Qualiclinic K ft, Budapest
  - Pest megyei Flór Ferenc Kórház, Reumatológia-és Fizioterápiás Osztály, Kistarcsa
  - VITAL MEDICAL CENTER (VITÁL-MEDICINA Kft.), Veszprém
- Barzilai Medical Center, Ashkelon, Israel
- Poland (20):
  - Geo Medical Sp. z.o.o Szpital Geo Medical, Katowice
  - Moja Przychodnia, Katowice
  - C.M. Silmedic Sp. z o.o., Katowice
  - Malopolskie Badania Kliniczne Sp. z o.o. s.k., Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne LUX MED, Krakow
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Szpital Uniwersytecki w Krakowie, Zaklad Radiologii, Krakow
  - Top Medical, Lublin
  - Zespol Poradni Specjalistycznych REUMED, Wallenroda Filia nr 1, Lublin
  - NZOZ JAMED Pracownia Rentgenowska Jerema Antoszewski, Poznan
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan
  - Klinika Alfa, Sochaczew
  - RCMed Oddzial Sochaczew, Sochaczew
  - Szpital Powiatowy w Sochaczewie, Sochaczew
  - Szpital Sw. Elzbiety, Mokotowskie Centrum Medyczne, Zaklad Diagnostyki, Warsaw
  - "Reumatika - Centrum Reumatologii" NZOZ, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Centrum Medyczne Medix, Wroclaw
- Russia (6):
  - Limited Liability Company Medical Center "Rheuma-Med", Kemerovo
  - State Budgetary Healthcare Institution "Orenburg Regional Clinical Hospital", Orenburg
  - Limited Liability Company "Sanavita", Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
  - RSBHI "Smolensk Regional Clinical Hospital", Smolensk
  - Limited Liability Company "BioMed", Vladimir
- South Korea (3):
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Hanyang University Seoul Hospital, Seoul
- Turkey (Türkiye) (8):
  - Ankara Universitesi Tip Fakultesi Ibn-i Sina Hastanesi, Ankara
  - Ankara Universitesi Tip Fakultesi, Ibn-i Sina Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ic Hastaliklari Anabilim, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi, Ic Hastaliklari, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Marmara Univ. Istanbul Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Izmir Katip Celebi Univ Ataturk Egitim ve Arastirma Hastanesi, Izmir
  - Izmir Katip Celebi Univ. Ataturk Egitim ve Arastirma Hastanesi, Izmir
- Ukraine (5):
  - Kyiv City Clinical Hospital # 3, Rheumatology Department, Kyiv
  - Lviv Communal Clinical Hospital #4, Rheumatology department, Lviv
  - Military-Medical Clinical Center (Clinical Hospital with 200 beds) of State Border Guard Service of, Lviv
  - Ternopil University Hospital, Department of Rheumatology,, Ternopil
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrohov, rheumatology department,, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Deodhar A, Akar S, Curtis JR, El-Zorkany B, Magrey M, Wang C, Wu J, Makgoeng SB, Vranic I, Menon S, Fleishaker DL, Diehl AM, Fallon L, Yndestad A, Landewe RBM. Integrated safety analysis of tofacitinib from Phase 2 and 3 trials of patients with ankylosing spondylitis. Adv Rheumatol. 2024 Dec 18;64(1):87. doi: 10.1186/s42358-024-00402-x. PMID 39695887
- [Derived] Gossec L, Walsh JA, Sengupta R, Bushmakin AG, Cappelleri JC, Yndestad A, Dina O, Cella D. Improvement of Fatigue in Patients with Ankylosing Spondylitis Receiving Tofacitinib: Analyses of a Phase 3 Randomized Controlled Trial. Rheumatol Ther. 2025 Feb;12(1):85-98. doi: 10.1007/s40744-024-00727-5. Epub 2024 Dec 13. PMID 39671076
- [Derived] Norton H, Sliwinska-Stanczyk P, Hala T, El-Zorkany B, Stockert L, Mundayat R, Wang L, Ritchlin CT. Tofacitinib Efficacy/Safety in Patients with Ankylosing Spondylitis by Baseline Body Mass Index: A Post Hoc Analysis of Phase 2/3 Trials. Rheumatol Ther. 2025 Feb;12(1):67-84. doi: 10.1007/s40744-024-00726-6. Epub 2024 Dec 5. PMID 39636343
- [Derived] Ogdie A, Kristensen LE, Soriano ER, Akar S, Sun Y, Gruben D, Fallon L, Kinch CD, Gladman DD. Efficacy and Safety of Tofacitinib in Patients with Psoriatic Arthritis or Ankylosing Spondylitis by Cigarette Smoking Status. Rheumatol Ther. 2024 Dec;11(6):1649-1664. doi: 10.1007/s40744-024-00711-z. Epub 2024 Sep 25. PMID 39320582
- [Derived] Deodhar A, Baraliakos X, Magrey M, Gensler LS, Thorat AV, Pemmaraju SK, Cadatal MJ, Nash P. Efficacy and Safety of Tofacitinib in Ankylosing Spondylitis by Baseline C-Reactive Protein Level: Post Hoc Analysis of Phase II and Phase III Clinical Trials. J Rheumatol. 2024 Aug 1;51(8):772-780. doi: 10.3899/jrheum.2023-1198. PMID 38825359
- [Derived] Navarro-Compan V, Deodhar A, Bahiri R, Bushmakin AG, Cappelleri JC, Rammaoui J. Time to improvement of pain, morning stiffness, fatigue, and disease activity in patients with ankylosing spondylitis treated with tofacitinib: a post hoc analysis. Arthritis Res Ther. 2024 May 24;26(1):105. doi: 10.1186/s13075-024-03313-w. PMID 38790040
- [Derived] Kristensen LE, Deodhar A, Leung YY, Vranic I, Mortezavi M, Fallon L, Yndestad A, Kinch CD, Gladman DD. Risk Stratification of Patients with Psoriatic Arthritis and Ankylosing Spondylitis for Treatment with Tofacitinib: A Review of Current Clinical Data. Rheumatol Ther. 2024 Jun;11(3):487-499. doi: 10.1007/s40744-024-00662-5. Epub 2024 May 2. PMID 38696034
- [Derived] Magrey M, Wei JC, Yndestad A, Bushmakin AG, Cappelleri JC, Dina O, Deodhar A. Relationships of Work Productivity and Activity Impairment With Patient-Reported Outcomes in Ankylosing Spondylitis: Results From Two Trials. Arthritis Care Res (Hoboken). 2024 Mar;76(3):359-365. doi: 10.1002/acr.25267. Epub 2024 Jan 5. PMID 37909386
- [Derived] Cella D, Lenderking WR, Chongpinitchai P, Bushmakin AG, Dina O, Wang L, Cappelleri JC, Navarro-Compan V. Functional Assessment of Chronic Illness Therapy-Fatigue is a reliable and valid measure in patients with active ankylosing spondylitis. J Patient Rep Outcomes. 2022 Sep 23;6(1):100. doi: 10.1186/s41687-022-00508-0. PMID 36138330
- [Derived] Navarro-Compan V, Wei JC, Van den Bosch F, Magrey M, Wang L, Fleishaker D, Cappelleri JC, Wang C, Wu J, Dina O, Fallon L, Strand V. Effect of tofacitinib on pain, fatigue, health-related quality of life and work productivity in patients with active ankylosing spondylitis: results from a phase III, randomised, double-blind, placebo-controlled trial. RMD Open. 2022 Jun;8(2):e002253. doi: 10.1136/rmdopen-2022-002253. PMID 35654457
- [Derived] Deodhar A, Sliwinska-Stanczyk P, Xu H, Baraliakos X, Gensler LS, Fleishaker D, Wang L, Wu J, Menon S, Wang C, Dina O, Fallon L, Kanik KS, van der Heijde D. Tofacitinib for the treatment of ankylosing spondylitis: a phase III, randomised, double-blind, placebo-controlled study. Ann Rheum Dis. 2021 Aug;80(8):1004-1013. doi: 10.1136/annrheumdis-2020-219601. Epub 2021 Apr 27. PMID 33906853
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921120

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety data was planned to be collected and reported for both: Week 0 to Week 16 and from Week 0 to Week 48.
Groups:
- Tofacitinib: Participants received Tofacitinib tablets 5 milligram (mg), twice daily for 48 weeks.
- Placebo Then Tofacitinib: Participants received tofacitinib matching placebo tablets, twice daily for 16 weeks followed by tofacitinib tablets 5 mg, twice daily for next 32 weeks (i.e. up to Week 48).
Period: Up to Week 16
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Started | 134 | 136
Treated | 133 | 136
Completed | 132 | 133
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Randomized, but not treated | 1 | 0
Period: Week 16 to Week 48
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Started | 132 | 133
Treated | 132 | 133
Completed | 125 | 127
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: included all participants who were randomized and received at least one dose of the investigational product (that is [i.e.], tofacitinib or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib | Placebo Then Tofacitinib | Total
Number analyzed (Participants) | 133 | 136 | 269
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (11.85) | 40.0 (11.06) | 41.1 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 28 | 45
  Male | 116 | 108 | 224
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 107 | 106 | 213
  Asian | 25 | 30 | 55
  Not reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Assessment of SpondyloArthritis International Society (ASAS)20 Response at Week 16
Description: ASAS20 assess 4 domains: Patient Global Assessment of Disease (PGA) (assess disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity), total back pain (scale of 0 [no pain] to 10 [most severe pain], high score=more severity), Function (Bath Ankylosing Spondylitis Functional Index [BASFI]; participant's level of ability on scale of 0 [easy] to 10 [impossible], low score= better functional health) and Inflammation (morning stiffness, Mean of Question [Q]5 and Q6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] defined as 6-item questionnaire measure disease activity on a scale of 0 [none] to 10 [severe], high score=more disease activity). ASAS20 response: greater than or equal to (>=) 20 percent (%) improvement from baseline in disease activity and absolute change of >=1 unit in >=3 domains and no worsening of >=20% and an absolute change of >=1 unit in remaining domain.
Time Frame: Week 16
Population: Full Analysis Set (FAS): included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Here, on-drug data was used and missing response (MR) was considered to be Non-response (NR) (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants | 56.39 | 29.41
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via Cochran-Mantel-Haenszel (CMH) approach; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 27.08, 95% CI 2-sided [15.89 to 38.28], Standard Error of Mean 5.71

2. Secondary Outcome: Percentage of Participants Achieving Ankylosing Spondylitis (ASAS)40 Response at Week 16
Description: ASAS40 assessed 4 domains: the "PGA" (assess disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity), total back pain (on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity), Function (from BASFI: assess participant's level of ability on a scale of 0 [easy] to 10 [impossible], lower scores= better functional health) and Inflammation (morning stiffness, Mean of Q5 and Q6 of BASDAI defined as 6 item questionnaire: measures disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity). ASAS40 response: >=40% and >=2 units improvement in >=3 domains and no worsening at all in the remaining domain.
Time Frame: Week 16
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Here, on-drug data was used and missing response (MR) was considered to be Non-response (NR) (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants | 40.60 | 12.50
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 28.17, 95% CI 2-sided [18.26 to 38.09], Standard Error of Mean 5.06

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily living (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Treatment-emergent were events between first dose of study drug and up to 48 weeks that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Week 16 and Baseline up to Week 48
Population: Safety analysis set: included all participants who were randomized and received at least one dose of the investigational product (i.e., tofacitinib or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Participants
  Up to Week 16 | 73 | 70
  Up to Week 48 | 103 | 93

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) by Severity
Description: AE: any untoward medical occurrence in subject who receive study drug without regard to possibility of causal relationship. Treatment-emergent AEs were events that occurred between first dose of study drug and up to 48 weeks that were absent before treatment or that worsened relative to pretreatment state. The severity grades (mild, moderate and severe) were defined as - mild: did not interfere with participant's usual function, moderate: Interfered to some extent with participant's usual function and severe: Interfered significantly with participant's usual function.
Time Frame: Baseline up to Week 16 and Baseline up to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Participants
  Up to Week 16: Mild | 53 | 52
  Up to Week 16: Moderate | 18 | 18
  Up to Week 16: Severe | 2 | 0
  Up to Week 48: Mild | 57 | 57
  Up to Week 48: Moderate | 40 | 36
  Up to Week 48: Severe | 6 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Hematology (Hemoglobin, Hematocrit, Erythrocyte, Lymphocyte/Leukocyte, Neutrophil/Leukocyte <0.8*Lower limit of normal (LLN), Reticulocyte >1.5*Upper limit of normal (ULN), Erythrocyte Mean Corpuscular Volume, Erythrocyte Mean Corpuscular Hemoglobin, Erythrocyte Mean Corpuscular HGB Concentration <0.9*LLN, >1.1*ULN, Reticulocyte/Erythrocyte, Leukocyte >1.5*ULN, Lymphocyte, Neutrophil <0.8*LLN and >1.2*ULN, Basophil, Basophil/Leukocyte, Eosinophil, Eosinophil/Leukocyte, Monocyte, Monocyte/Leukocyte >1.2*ULN); Clinical Chemistry (Bilirubin, Glucose >1.5*ULN, AST, ALT, Gamma Glutamyl Transferase >3.0*ULN, Urea, Creatinine, Triglyceride, Cholesterol >1.3*ULN, LDL Cholesterol>1.2*ULN, Potassium, C Reactive Protein >1.1*ULN, Bicarbonate <0.9*LLN, Creatine Kinase >2.0*ULN, HDL Cholesterol <0.8*LLN), Urinalysis (Specific Gravity >1.035, pH >8, Glucose, Ketones, Protein, Hemoglobin >=1, Erythrocyte, Leukocyte >=20, Granular Cast, Hyaline Cast>1.
Time Frame: Baseline up to Week 16 and Baseline up to Week 48
Population: Safety analysis set: included all participants who were randomized and received at least one dose of the investigational product (i.e., tofacitinib or placebo). Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Participants
  Up to Week 16 | 106 | 129
  Up to Week 48 | 126 | 131

6. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for abnormalities in vital signs: Pulse rate <40 beats per minute (bpm) to >120 bpm, Sitting Diastolic blood pressure < 50 millimeter of mercury (mmHg), increase and decrease in change from baseline of >= 20mmHg, sitting systolic blood pressure < 90 mmHg, increase and decrease in change from baseline of >= 30mmHg.
Time Frame: Baseline up to Week 16 and Baseline up to Week 48
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Participants
  Up to Week 16, Pulse rate: <40 bpm | 0 | 0
  Up to Week 16, Pulse rate: >120 bpm | 0 | 0
  Up to Week 16, Sitting diastolic blood pressure: <50 mmHg | 0 | 0
  Up to Week 16, Sitting diastolic blood pressure: Change >= 20mmHg increase | 2 | 4
  Up to Week 16, Sitting diastolic blood pressure: Change >= 20mmHg decrease | 6 | 4
  Up to Week 16, Sitting systolic blood pressure: <90mmHg | 1 | 0
  Up to Week 16, Sitting systolic blood pressure: Change >= 30mmHg increase | 2 | 4
  Up to Week 16, Sitting systolic blood pressure: Change >= 30mmHg decrease | 2 | 5
  Up to Week 48, Pulse rate: <40 bpm | 0 | 0
  Up to Week 48, Pulse rate: >120 bpm | 0 | 1
  Up to Week 48, Sitting diastolic blood pressure: <50 mmHg | 0 | 0
  Up to Week 48, Sitting diastolic blood pressure: Change >= 20mmHg increase | 5 | 8
  Up to Week 48, Sitting diastolic blood pressure: Change >= 20mmHg decrease | 11 | 8
  Up to Week 48, Sitting systolic blood pressure: <90mmHg | 1 | 0
  Up to Week 48, Sitting systolic blood pressure: Change >= 30mmHg increase | 5 | 5
  Up to Week 48, Sitting systolic blood pressure: Change >= 30mmHg decrease | 5 | 7

7. Secondary Outcome: Number of Participants With Abnormalities in Physical Examination
Description: Complete physical examination: included general appearance, skin (presence of rash), heent (head, eyes, ears, nose and throat), lungs (auscultation), heart (auscultation for presence of murmurs, gallops, rubs), lower extremities (presence of peripheral edema), abdominal (palpation and auscultation), neurologic (mental status, station, gait, reflexes, motor and sensory function, coordination) and lymph nodes. Abnormalities in physical examination was based on investigator's discretion/clinical judgement.
Time Frame: Screening, Week 16, and Week 48
Population: Safety analysis set: included all participants who were randomized and received at least one dose of the investigational product (i.e., tofacitinib or placebo). Here, "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Participants
  Abdomen: Screening: number analyzed (Participants) | 133 | 135
  Abdomen: Screening | 2 | 1
  Abdomen: Week 16: number analyzed (Participants) | 132 | 132
  Abdomen: Week 16 | 1 | 2
  Abdomen: Week 48: number analyzed (Participants) | 119 | 119
  Abdomen: Week 48 | 1 | 1
  Extremities: Screening | 17 | 15
  Extremities: Week 16: number analyzed (Participants) | 132 | 132
  Extremities: Week 16 | 8 | 14
  Extremities: Week 48: number analyzed (Participants) | 119 | 119
  Extremities: Week 48 | 4 | 7
  General appearance: Screening: number analyzed (Participants) | 133 | 135
  General appearance: Screening | 10 | 11
  General appearance: Week 16: number analyzed (Participants) | 132 | 132
  General appearance: Week 16 | 9 | 9
  General appearance: Week 48: number analyzed (Participants) | 119 | 119
  General appearance: Week 48 | 7 | 6
  Head, eyes, ears, nose, throat: Screening: number analyzed (Participants) | 133 | 135
  Head, eyes, ears, nose, throat: Screening | 5 | 7
  Head, eyes, ears, nose, throat: Week 16: number analyzed (Participants) | 132 | 132
  Head, eyes, ears, nose, throat: Week 16 | 4 | 7
  Head, eyes, ears, nose, throat: Week 48: number analyzed (Participants) | 119 | 119
  Head, eyes, ears, nose, throat: Week 48 | 3 | 7
  Heart: Screening | 2 | 2
  Heart: Week 16: number analyzed (Participants) | 132 | 132
  Heart: Week 16 | 0 | 2
  Heart: Week 48: number analyzed (Participants) | 119 | 119
  Heart: Week 48 | 0 | 2
  Lungs: Screening | 1 | 0
  Lungs: Week 16: number analyzed (Participants) | 132 | 132
  Lungs: Week 16 | 0 | 0
  Lungs: Week 48: number analyzed (Participants) | 119 | 119
  Lungs: Week 48 | 0 | 0
  Lymph nodes: Screening | 2 | 3
  Lymph nodes: Week 16: number analyzed (Participants) | 132 | 131
  Lymph nodes: Week 16 | 1 | 2
  Lymph nodes: Week 48: number analyzed (Participants) | 119 | 119
  Lymph nodes: Week 48 | 1 | 2
  Neurological: Screening: number analyzed (Participants) | 133 | 135
  Neurological: Screening | 4 | 0
  Neurological: Week 16: number analyzed (Participants) | 132 | 131
  Neurological: Week 16 | 1 | 0
  Neurological: Week 48: number analyzed (Participants) | 119 | 119
  Neurological: Week 48 | 2 | 0
  Skin: Screening: number analyzed (Participants) | 133 | 135
  Skin: Screening | 18 | 18
  Skin: Week 16: number analyzed (Participants) | 132 | 132
  Skin: Week 16 | 14 | 13
  Skin: Week 48: number analyzed (Participants) | 119 | 119
  Skin: Week 48 | 12 | 12

8. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Twelve-lead electrocardiograms (ECGs) were obtained for all participants. Criteria for ECG abnormality: PR interval >=300 and a percent change from baseline of >=25 or 50%; QRS duration >=140 and a percent change from baseline of >=50%; QT interval >=500; QTCB, QTCF interval <480 or >=450, <500 or >=480, >=500, change from baseline of <60 and >=30, and change from baseline of >=60.
Time Frame: Baseline up to Week 16, Baseline up to Week 48
Population: Safety analysis set: included all participants who were randomized and received at least one dose of the investigational product (i.e., tofacitinib or placebo). Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 131 | 133
Participants
  Up to Week 16, PR interval: >=300: number analyzed (Participants) | 131 | 131
  Up to Week 16, PR interval: >=300 | 0 | 0
  Up to Week 16, PR interval: %Change>=25/50%: number analyzed (Participants) | 131 | 131
  Up to Week 16, PR interval: %Change>=25/50% | 0 | 1
  Up to Week 16, QRS duration: >=140: number analyzed (Participants) | 131 | 131
  Up to Week 16, QRS duration: >=140 | 1 | 1
  Up to Week 16, QRS duration: %Change>=50%: number analyzed (Participants) | 131 | 131
  Up to Week 16, QRS duration: %Change>=50% | 0 | 0
  Up to Week 16, QT interval: >=500: number analyzed (Participants) | 131 | 131
  Up to Week 16, QT interval: >=500 | 0 | 0
  Up to Week 16, QTCB interval: >=450 and <480: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCB interval: >=450 and <480 | 3 | 7
  Up to Week 16, QTCB interval: >=480 and <500: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCB interval: >=480 and <500 | 0 | 1
  Up to Week 16, QTCB interval: >=500: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCB interval: >=500 | 0 | 0
  Up to Week 16, QTCB interval: change >=30 and <60: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCB interval: change >=30 and <60 | 9 | 7
  Up to Week 16, QTCB interval: change >=60: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCB interval: change >=60 | 0 | 0
  Up to Week 16, QTCF interval: >=450 and <480: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCF interval: >=450 and <480 | 3 | 4
  Up to Week 16, QTCF interval: >=480 and <500: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCF interval: >=480 and <500 | 0 | 0
  Up to Week 16, QTCF interval: >=500: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCF interval: >=500 | 0 | 0
  Up to Week 16, QTCF interval: change >=30 and <60: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCF interval: change >=30 and <60 | 5 | 3
  Up to Week 16, QTCF interval: change >=60: number analyzed (Participants) | 131 | 131
  Up to Week 16, QTCF interval: change >=60 | 0 | 0
  Up to Week 48, PR interval: >=300 | 0 | 0
  Up to Week 48, PR interval: %Change>=25/50% | 0 | 1
  Up to Week 48, QRS duration: >=140 | 3 | 1
  Up to Week 48, QRS duration: %Change>=50% | 0 | 0
  Up to Week 48, QT interval: >=500 | 0 | 1
  Up to Week 48, QTCB interval: >=450 and <480 | 10 | 10
  Up to Week 48, QTCB interval: >=480 and <500 | 1 | 1
  Up to Week 48, QTCB interval: >=500 | 0 | 0
  Up to Week 48, QTCB interval: change >=30 and <60 | 14 | 11
  Up to Week 48, QTCB interval: change >=60 | 1 | 0
  Up to Week 48, QTCF interval: >=450 and <480 | 5 | 5
  Up to Week 48, QTCF interval: >=480 and <500 | 1 | 0
  Up to Week 48, QTCF interval: >=500 | 0 | 0
  Up to Week 48, QTCF interval: change >=30 and <60 | 9 | 7
  Up to Week 48, QTCF interval: change >=60 | 1 | 0

9. Secondary Outcome: Percentage of Participants Achieving ASAS20 Response at Weeks 2, 4, 8, 12, 24, 32, 40 and 48
Description: ASAS20 assess 4 domains: PGA of Disease (assess disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity), total back pain (scale of 0 [no pain] to 10 [most severe pain], high score=more severity), Function (BASFI; participant's level of ability on scale of 0 [easy] to 10 [impossible], low score= better functional health) and Inflammation (morning stiffness, Mean of Q5 and Q6 of BASDAI defined as 6-item questionnaire measure disease activity on a scale of 0 [none] to 10 [severe], high score=more disease activity). ASAS20 response: >= 20% improvement from baseline in disease activity and absolute change of >=1 unit in >=3 domains and no worsening of >=20% and an absolute change of >=1 unit in remaining domain.
Time Frame: Weeks 2, 4, 8, 12, 24, 32, 40 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants
  Week 2 | 28.57 | 10.29
  Week 4 | 51.13 | 19.85
  Week 8 | 57.14 | 25.00
  Week 12 | 63.91 | 29.41
  Week 24 | 63.16 | 59.56
  Week 32 | 68.42 | 64.71
  Week 40 | 68.42 | 66.91
  Week 48 | 65.41 | 60.29
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 2: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 18.28, 95% CI 2-sided [9.06 to 27.50], Standard Error of Mean 4.70
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 4: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 31.35, 95% CI 2-sided [20.64 to 42.06], Standard Error of Mean 5.47
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 8: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 32.24, 95% CI 2-sided [21.32 to 43.17], Standard Error of Mean 5.57
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 12: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 34.61, 95% CI 2-sided [23.63 to 45.58], Standard Error of Mean 5.60
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 24: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p = 0.5360, Cochran-Mantel-Haenszel; Difference in percentage = 3.65, 95% CI 2-sided [-7.92 to 15.22], Standard Error of Mean 5.90
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 32: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p = 0.4971, Cochran-Mantel-Haenszel; Difference in percentage = 3.83, 95% CI 2-sided [-7.22 to 14.87], Standard Error of Mean 5.63
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 40: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p = 0.7792, Cochran-Mantel-Haenszel; Difference in percentage = 1.58, 95% CI 2-sided [-9.49 to 12.66], Standard Error of Mean 5.65
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p = 0.3685, Cochran-Mantel-Haenszel; Difference in percentage = 5.22, 95% CI 2-sided [-6.15 to 16.58], Standard Error of Mean 5.80

10. Secondary Outcome: Percentage of Participants Achieving ASAS40 Response at Weeks 2, 4, 8, 12, 24, 32, 40 and 48
Description: as for outcome 2
Time Frame: Weeks 2, 4, 8, 12, 24, 32, 40 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants
  Week 2 | 10.53 | 4.41
  Week 4 | 27.07 | 3.68
  Week 8 | 34.59 | 5.88
  Week 12 | 42.86 | 11.76
  Week 24 | 48.12 | 41.91
  Week 32 | 50.38 | 44.12
  Week 40 | 50.38 | 42.65
  Week 48 | 50.38 | 44.85
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0548, Cochran-Mantel-Haenszel; Difference in percentage = 6.12, 95% CI 2-sided [-0.13 to 12.37], Standard Error of Mean 3.19
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 23.43, 95% CI 2-sided [15.30 to 31.56], Standard Error of Mean 4.15
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 28.56, 95% CI 2-sided [19.66 to 37.47], Standard Error of Mean 4.54
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 31.18, 95% CI 2-sided [21.34 to 41.02], Standard Error of Mean 5.02
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.2926, Cochran-Mantel-Haenszel; Difference in percentage = 6.29, 95% CI 2-sided [-5.43 to 18.01], Standard Error of Mean 5.98
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.2856, Cochran-Mantel-Haenszel; Difference in percentage = 6.37, 95% CI 2-sided [-5.32 to 18.06], Standard Error of Mean 5.97
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.1894, Cochran-Mantel-Haenszel; Difference in percentage = 7.83, 95% CI 2-sided [-3.87 to 19.54], Standard Error of Mean 5.97
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.3544, Cochran-Mantel-Haenszel; Difference in percentage = 5.59, 95% CI 2-sided [-6.24 to 17.43], Standard Error of Mean 6.04

11. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score Using C-Reactive Protein (ASDAS[CRP]) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: ASDAS(CRP) was derived using BASDAI (6-item questionnaire measures disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and PGA (measure disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity) and calculated by using the following formula, 0.121 x Back Pain (Q2 of BASDAI) + 0.058 x Duration of Morning Stiffness (Q6 of BASDAI) + 0.110 x PGA + 0.073 x Peripheral Pain/Swelling (Q3 of BASDAI) + 0.579 x Ln(high sensitivity [hs] CRP mg/Liter [L] + 1). If hsCRP values were smaller than 2 mg/L, they were set to 2 mg/L in the formula. The range of score was >= 0.636 to no defined upper limit. A negative change from baseline value indicates decrease in disease activity; a positive change from baseline value indicates increase in disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: Full Analysis Set (FAS): included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Here, on-drug data was used and missing response was not imputed. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -0.88 (0.056) | -0.17 (0.056)
  Week 4 | -1.14 (0.065) | -0.24 (0.065)
  Week 8 | -1.30 (0.074) | -0.24 (0.074)
  Week 12 | -1.38 (0.075) | -0.28 (0.075)
  Week 16 | -1.36 (0.073) | -0.39 (0.073)
  Week 24 | -1.51 (0.082) | -1.32 (0.081)
  Week 32 | -1.56 (0.084) | -1.37 (0.084)
  Week 40 | -1.65 (0.086) | -1.40 (0.086)
  week 48 | -1.70 (0.087) | -1.50 (0.086)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 2: Analysis performed using Mixed model for repeated measures (MMRM) which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.71, 95% CI 2-sided [-0.85 to -0.57], Standard Error of Mean 0.072
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 4: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.90, 95% CI 2-sided [-1.07 to -0.74], Standard Error of Mean 0.083
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 8: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.06, 95% CI 2-sided [-1.25 to -0.87], Standard Error of Mean 0.095
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 12: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.09, 95% CI 2-sided [-1.28 to -0.90], Standard Error of Mean 0.096
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.98, 95% CI 2-sided [-1.16 to -0.79], Standard Error of Mean 0.093
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 24: Analysis performed using Mixed model for repeated measures (MMRM) which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.0623, Mixed Models Analysis; LS mean difference = -0.19, 95% CI 2-sided [-0.40 to 0.01], Standard Error of Mean 0.103
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 32: Analysis performed using Mixed model for repeated measures (MMRM) which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.0836, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-0.39 to 0.02], Standard Error of Mean 0.106
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 40: Analysis performed using Mixed model for repeated measures (MMRM) which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.0205, Mixed Models Analysis; LS mean difference = -0.25, 95% CI 2-sided [-0.47 to -0.04], Standard Error of Mean 0.108
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48: Analysis performed using Mixed model for repeated measures (MMRM) which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.0614, Mixed Models Analysis; LS mean difference = -0.20, 95% CI 2-sided [-0.42 to 0.01], Standard Error of Mean 0.108

12. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Blood samples were collected for analysis of hsCRP using an assay analyzed by central laboratory. hsCRP is an acute phase reactant, which was indicative of inflammation and of its severity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Here, on-drug data was used and missing response was not imputed. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Milligrams per deciliter (mg/dL)
  Week 2 | -1.07 (0.089) | -0.14 (0.088)
  Week 4 | -1.06 (0.094) | -0.14 (0.094)
  Week 8 | -1.05 (0.153) | -0.03 (0.152)
  Week 12 | -1.11 (0.089) | -0.15 (0.090)
  Week 16 | -1.05 (0.096) | -0.09 (0.096)
  Week 24 | -1.21 (0.058) | -1.16 (0.058)
  Week 32 | -1.16 (0.076) | -1.08 (0.075)
  Week 40 | -1.22 (0.089) | -1.09 (0.089)
  Week 48 | -1.17 (0.081) | -1.11 (0.080)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 2: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.93, 95% CI 2-sided [-1.15 to -0.70], Standard Error of Mean 0.113
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.92, 95% CI 2-sided [-1.16 to -0.68], Standard Error of Mean 0.121
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.02, 95% CI 2-sided [-1.40 to -0.63], Standard Error of Mean 0.196
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.96, 95% CI 2-sided [-1.19 to -0.74], Standard Error of Mean 0.115
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.96, 95% CI 2-sided [-1.20 to -0.72], Standard Error of Mean 0.122
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 24: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.4731, Mixed Models Analysis; LS mean difference = -0.05, 95% CI 2-sided [-0.20 to 0.09], Standard Error of Mean 0.073
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 32: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.4055, Mixed Models Analysis; LS mean difference = -0.08, 95% CI 2-sided [-0.26 to 0.11], Standard Error of Mean 0.094
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 40: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.2648, Mixed Models Analysis; LS mean difference = -0.12, 95% CI 2-sided [-0.34 to 0.09], Standard Error of Mean 0.111
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.5558, Mixed Models Analysis; LS mean difference = -0.06, 95% CI 2-sided [-0.25 to 0.14], Standard Error of Mean 0.099

13. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score at Weeks 16 and 48
Description: The ASQoL was an 18-item questionnaire assessed the amount of restriction participant experienced in daily activities, level of pain and fatigue, and the impact on the participant's emotional state. Each item was scored as 0 (no impact) or 1 (yes - impact). A total score was calculated by summing the items. The total score ranged from 0 (no impact) to 18 (yes-impact), with higher values indicated more impaired health-related quality of life.
Time Frame: Baseline, Weeks 16 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Here, on-drug data was used and missing response was not imputed. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Here, "number analyzed" signifies participants evaluable for this outcome measure for specified time point.
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 129 | 131
Units on scale
  Week 16: number analyzed (Participants) | 129 | 130
  Week 16 | -4.03 (0.404) | -2.01 (0.405)
  Week 48 | -5.97 (0.454) | -4.70 (0.451)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16: Analysis performed using Analysis of covariance (ANCOVA) model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.0001, ANCOVA; LS mean difference = -2.02, 95% CI 2-sided [-3.03 to -1.01], Standard Error of Mean 0.513
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0270, Mixed Models Analysis; LS mean difference = -1.26, 95% CI 2-sided [-2.38 to -0.14], Standard Error of Mean 0.567

14. Secondary Outcome: Change From Baseline in Short-Form-36 Health Survey-Version 2 Acute (SF-36v2) Score at Weeks 16 and 48
Description: SF-36 v.2 (Acute): 36-item generic health status measure. It measured 8 general health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, mental health. These domains were aggregated into 2 summary scores - physical component summary (PCS), mental component summary (MCS). Four domains comprised PCS score (physical functioning, role-physical, bodily pain, general health) and remaining 4 domains comprised MCS score (vitality, social functioning, role-emotional, mental health). Normalized domain scores, PCS, MCS scores are used in analyses. Component and domain scores were scored by using United States 1998 general population norm. Resulting norm-based T-scores for both the SF36 version 2 and SF36 health domain scale and component summary measures had means of 50 and standard deviations of 10. Higher PCS/MCS/domain score represent better health status.
Time Frame: Baseline, Weeks 16 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 129 | 130
Units on a scale
  Week 16: Physical Functioning | 5.52 (0.665) | 3.29 (0.665)
  Week 16: Role-Physical | 6.13 (0.744) | 3.13 (0.745)
  Week 16: Bodily Pain | 7.93 (0.710) | 3.47 (0.713)
  Week 16: General Health | 5.00 (0.617) | 1.76 (0.618)
  Week 16: Vitality | 5.34 (0.864) | 3.56 (0.869)
  Week 16: Social Functioning | 5.45 (0.835) | 2.49 (0.837)
  Week 16: Role-Emotional | 4.13 (1.020) | 2.05 (1.017)
  Week 16: Mental Health | 3.57 (0.886) | 2.49 (0.888)
  Week 16: Physical Component Summary | 6.69 (0.588) | 3.14 (0.590)
  Week 16: Mental Component Summary | 3.45 (0.914) | 2.13 (0.915)
  Week 48: Physical Functioning | 7.80 (0.775) | 6.94 (0.766)
  Week 48: Role-Physical | 8.66 (0.870) | 7.29 (0.862)
  Week 48: Bodily Pain | 11.67 (0.920) | 9.55 (0.912)
  Week 48: General Health | 6.31 (0.777) | 5.10 (0.770)
  Week 48: Vitality | 9.83 (0.997) | 9.28 (0.992)
  Week 48: Social Functioning | 8.16 (0.923) | 6.77 (0.915)
  Week 48: Role-Emotional | 7.17 (1.004) | 6.32 (0.989)
  Week 48: Mental Health | 7.10 (0.960) | 6.45 (0.954)
  Week 48: Physical Component Summary | 8.81 (0.720) | 7.39 (0.714)
  Week 48: Mental Component Summary | 7.07 (0.926) | 6.35 (0.920)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Physical Functioning: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.0088, ANCOVA; LS mean difference = 2.22, 95% CI 2-sided [0.56 to 3.88], Standard Error of Mean 0.841
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Role-Physical: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.0016, ANCOVA; LS mean difference = 3.00, 95% CI 2-sided [1.15 to 4.85], Standard Error of Mean 0.939
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Bodily Pain: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 4.46, 95% CI 2-sided [2.69 to 6.23], Standard Error of Mean 0.900
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, General Health: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 3.24, 95% CI 2-sided [1.70 to 4.78], Standard Error of Mean 0.781
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Vitality: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.1065, ANCOVA; LS mean difference = 1.78, 95% CI 2-sided [-0.38 to 3.94], Standard Error of Mean 1.098
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Social Functioning: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.0055, ANCOVA; LS mean difference = 2.96, 95% CI 2-sided [0.88 to 5.05], Standard Error of Mean 1.059
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Role-Emotional: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.1084, ANCOVA; LS mean difference = 2.08, 95% CI 2-sided [-0.46 to 4.61], Standard Error of Mean 1.289
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Mental Health: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.3379, ANCOVA; LS mean difference = 1.08, 95% CI 2-sided [-1.13 to 3.29], Standard Error of Mean 1.124
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Physical Component Summary: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 3.55, 95% CI 2-sided [2.09 to 5.02], Standard Error of Mean 0.744
Statistical Analysis 10: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Mental Component Summary: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.2529, ANCOVA; LS mean difference = 1.33, 95% CI 2-sided [-0.95 to 3.61], Standard Error of Mean 1.158
Statistical Analysis 11: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Physical Functioning: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.3744, Mixed Models Analysis; LS mean difference = 0.86, 95% CI 2-sided [-1.04 to 2.76], Standard Error of Mean 0.964
Statistical Analysis 12: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Role-Physical: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.2091, Mixed Models Analysis; LS mean difference = 1.36, 95% CI 2-sided [-0.77 to 3.50], Standard Error of Mean 1.083
Statistical Analysis 13: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Bodily Pain: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.0654, Mixed Models Analysis; LS mean difference = 2.12, 95% CI 2-sided [-0.14 to 4.38], Standard Error of Mean 1.146
Statistical Analysis 14: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, General Health: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.2100, Mixed Models Analysis; LS mean difference = 1.22, 95% CI 2-sided [-0.69 to 3.12], Standard Error of Mean 0.968
Statistical Analysis 15: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Vitality: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.6568, Mixed Models Analysis; LS mean difference = 0.56, 95% CI 2-sided [-1.90 to 3.01], Standard Error of Mean 1.248
Statistical Analysis 16: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Social Functioning: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.2288, Mixed Models Analysis; LS mean difference = 1.39, 95% CI 2-sided [-0.88 to 3.66], Standard Error of Mean 1.152
Statistical Analysis 17: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Role-Emotional: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.4955, Mixed Models Analysis; LS mean difference = 0.85, 95% CI 2-sided [-1.61 to 3.32], Standard Error of Mean 1.250
Statistical Analysis 18: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Mental Health: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.5888, Mixed Models Analysis; LS mean difference = 0.65, 95% CI 2-sided [-1.71 to 3.01], Standard Error of Mean 1.200
Statistical Analysis 19: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Physical Component Summary: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.1150, Mixed Models Analysis; LS mean difference = 1.42, 95% CI 2-sided [-0.35 to 3.18], Standard Error of Mean 0.896
Statistical Analysis 20: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Mental Component Summary: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.5347, Mixed Models Analysis; LS mean difference = 0.72, 95% CI 2-sided [-1.56 to 3.00], Standard Error of Mean 1.158

15. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Scores: Cervical Rotation Angle at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASMI assess axial status and spinal mobility. It composed of 5 clinical measures: lateral spinal flexion, tragus-to-wall distance, lumbar flexion (modified Schober), maximal intermalleolar distance, cervical rotation. BASMI - Linear Method score was average of 5 individual component score mapped between 0 and 10, high score=more impairment of axial status, spinal mobility. For cervical rotation angle, participant sit straight on chair with chin level and hands on knees. Blinded assessor place goniometer at top of head in line with nose and ask participant to rotate neck maximally to left, follows with goniometer and record angle between sagittal plane and new plane after rotation. A second reading obtained and both readings recorded. Procedure repeated for right side. Better of two for each side was selected for scoring. Scoring done by calculating mean of left and right measurement and recorded in degrees (range: 0 to 90), higher cervical rotation value=better health status.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Degrees
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Degrees
  Week 2 | 2.25 (0.701) | 0.95 (0.698)
  Week 4 | 3.63 (0.797) | 2.07 (0.792)
  Week 8 | 6.26 (0.825) | 2.44 (0.824)
  Week 12 | 6.24 (1.002) | 2.92 (1.004)
  Week 16 | 7.74 (1.009) | 3.00 (1.008)
  Week 24 | 7.68 (1.139) | 7.49 (1.131)
  Week 32 | 7.25 (1.087) | 8.23 (1.080)
  Week 40 | 7.62 (1.215) | 8.34 (1.207)
  Week 48 | 7.63 (1.201) | 8.23 (1.188)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.1513, Mixed Models Analysis; LS mean difference = 1.29, 95% CI 2-sided [-0.48 to 3.06], Standard Error of Mean 0.898
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.1279, Mixed Models Analysis; LS mean difference = 1.56, 95% CI 2-sided [-0.45 to 3.56], Standard Error of Mean 1.020
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LS mean difference = 3.83, 95% CI 2-sided [1.75 to 5.90], Standard Error of Mean 1.056
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.0102, Mixed Models Analysis; LS mean difference = 3.32, 95% CI 2-sided [0.79 to 5.84], Standard Error of Mean 1.282
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LS mean difference = 4.73, 95% CI 2-sided [2.20 to 7.26], Standard Error of Mean 1.285
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.8950, Mixed Models Analysis; LS mean difference = 0.19, 95% CI 2-sided [-2.64 to 3.02], Standard Error of Mean 1.439
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.4732, Mixed Models Analysis; LS mean difference = -0.98, 95% CI 2-sided [-3.67 to 1.71], Standard Error of Mean 1.365
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.6359, Mixed Models Analysis; LS mean difference = -0.72, 95% CI 2-sided [-3.72 to 2.28], Standard Error of Mean 1.523
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.6894, Mixed Models Analysis; LS mean difference = -0.60, 95% CI 2-sided [-3.54 to 2.35], Standard Error of Mean 1.495

16. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Scores: Intermalleolar Distance at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASMI assessed axial status and spinal mobility, using linear function. It composed of 5 clinical measures: lateral spinal flexion, tragus-to-wall distance, lumbar flexion (modified Schober), maximal intermalleolar distance, cervical rotation. BASMI - Linear Method score was average of 5 individual component scores mapped between 0 and 10, with higher scores indicating more impairment of axial status and spinal mobility. For the assessment of intermalleolar distances, participant should lie supine with the knees straight and feet/toes pointing straight up and asked to separate the legs as far as possible and the distance between the medial malleoli was measured (in Centimeters [cm] to the nearest 0.1 cm). Distance (in cm) was greater than or equal to 0, with no maximum defined range: higher intermalleolar distance value indicates better health status.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Centimeters
  Week 2 | 2.29 (0.733) | 0.90 (0.730)
  Week 4 | 3.62 (0.861) | 0.84 (0.856)
  Week 8 | 4.68 (0.979) | 1.36 (0.976)
  Week 12 | 5.33 (1.106) | 1.97 (1.108)
  Week 16 | 6.84 (1.084) | 2.64 (1.082)
  Week 24 | 7.79 (1.177) | 4.39 (1.174)
  Week 32 | 8.98 (1.221) | 5.32 (1.215)
  Week 40 | 8.60 (1.229) | 4.75 (1.222)
  Week 48 | 7.83 (1.233) | 4.34 (1.222)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.1410, Mixed Models Analysis; LS mean difference = 1.39, 95% CI 2-sided [-0.46 to 3.24], Standard Error of Mean 0.940
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0122, Mixed Models Analysis; LS mean difference = 2.78, 95% CI 2-sided [0.61 to 4.95], Standard Error of Mean 1.102
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0085, Mixed Models Analysis; LS mean difference = 3.32, 95% CI 2-sided [0.86 to 5.79], Standard Error of Mean 1.252
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.0184, Mixed Models Analysis; LS mean difference = 3.36, 95% CI 2-sided [0.57 to 6.15], Standard Error of Mean 1.416
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0026, Mixed Models Analysis; LS mean difference = 4.19, 95% CI 2-sided [1.47 to 6.91], Standard Error of Mean 1.380
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0236, Mixed Models Analysis; LS mean difference = 3.40, 95% CI 2-sided [0.46 to 6.35], Standard Error of Mean 1.495
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0182, Mixed Models Analysis; LS mean difference = 3.66, 95% CI 2-sided [0.63 to 6.70], Standard Error of Mean 1.541
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0133, Mixed Models Analysis; LS mean difference = 3.85, 95% CI 2-sided [0.81 to 6.90], Standard Error of Mean 1.545
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0245, Mixed Models Analysis; LS mean difference = 3.49, 95% CI 2-sided [0.45 to 6.52], Standard Error of Mean 1.541

17. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Scores: Lateral Spinal Flexion at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASMI assess axial status, spinal mobility, using linear function. It composed of 5 clinical measures. BASMI - Linear Method score-average of 5 component scores mapped between 0 and 10, with high scores =more impairment of axial status, spinal mobility. For assessment of lateral spinal flexion: participant stand upright with head and back rest against wall as close as possible with shoulders level and feet 30 cm apart and feet parallel. At tip of middle finger, place a mark on thigh. This neutral position recorded. Participant bend sideways without bending knees or lifting heels while attempting to keep shoulders in same position (flexion position). Second mark placed, lateral flexion recorded (left or right as appropriate) using cm tape measure. Two tries for left, two tries for right measured. Result of two tries recorded for left and right separately in cm to nearest 0.1 cm. Distance (in cm) should be >=0, with no maximum defined range: high value indicates better health status.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Centimeters
  Week 2 | 0.60 (0.200) | -0.21 (0.199)
  Week 4 | 0.96 (0.235) | -0.10 (0.233)
  Week 8 | 1.34 (0.238) | 0.15 (0.237)
  Week 12 | 1.42 (0.214) | -0.21 (0.214)
  Week 16 | 1.79 (0.269) | -0.08 (0.269)
  Week 24 | 1.70 (0.278) | 0.75 (0.276)
  Week 32 | 1.90 (0.319) | 1.31 (0.316)
  Week 40 | 2.15 (0.332) | 1.37 (0.329)
  Week 48 | 1.64 (0.345) | 1.34 (0.340)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0018, Mixed Models Analysis; LS mean difference = 0.81, 95% CI 2-sided [0.30 to 1.32], Standard Error of Mean 0.257
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0005, Mixed Models Analysis; LS mean difference = 1.06, 95% CI 2-sided [0.47 to 1.65], Standard Error of Mean 0.301
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LS mean difference = 1.19, 95% CI 2-sided [0.59 to 1.79], Standard Error of Mean 0.305
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 1.63, 95% CI 2-sided [1.09 to 2.17], Standard Error of Mean 0.274
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 1.87, 95% CI 2-sided [1.20 to 2.55], Standard Error of Mean 0.344
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0075, Mixed Models Analysis; LS mean difference = 0.95, 95% CI 2-sided [0.26 to 1.65], Standard Error of Mean 0.353
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.1489, Mixed Models Analysis; LS mean difference = 0.58, 95% CI 2-sided [-0.21 to 1.38], Standard Error of Mean 0.403
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0609, Mixed Models Analysis; LS mean difference = 0.78, 95% CI 2-sided [-0.04 to 1.61], Standard Error of Mean 0.417
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.4822, Mixed Models Analysis; LS mean difference = 0.30, 95% CI 2-sided [-0.54 to 1.15], Standard Error of Mean 0.429

18. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Scores: Lumbar Flexion (Modified Schober) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASMI assessed axial status and spinal mobility. BASMI - Linear Method score was average of 5 individual component scores mapped between 0 and 10, with higher scores indicating more impairment of axial status and spinal mobility. For the assessment of lumbar flexion, With the participant standing erect and outer edges of feet 30 cm apart, a mark was placed in the midpoint of a line that joins the posterior superior iliac spines (baseline mark). A second mark (A) was placed 10 cm above the baseline mark and a third mark (B) 5 cm below the baseline mark. Then have the participant maximally bend forward, keeping the knees fully extended. With the participant's spine in full flexion, the distance between marks A and B (in cm to the nearest 0.1 cm) was re-measured. Distance (in cm) was greater than or equal to 0, with no maximum defined range. Higher value indicates better health status.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Centimeters
  Week 2 | 0.30 (0.102) | -0.07 (0.102)
  Week 4 | 0.41 (0.102) | -0.11 (0.102)
  Week 8 | 0.32 (0.116) | -0.17 (0.115)
  Week 12 | 0.26 (0.111) | -0.22 (0.111)
  Week 16 | 0.46 (0.115) | -0.06 (0.115)
  Week 24 | 0.51 (0.149) | 0.20 (0.148)
  Week 32 | 0.64 (0.143) | 0.39 (0.142)
  Week 40 | 0.58 (0.156) | 0.50 (0.155)
  Week 48 | 0.45 (0.146) | 0.35 (0.144)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0047, Mixed Models Analysis; LS mean difference = 0.37, 95% CI 2-sided [0.12 to 0.63], Standard Error of Mean 0.131
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LS mean difference = 0.52, 95% CI 2-sided [0.26 to 0.77], Standard Error of Mean 0.131
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0012, Mixed Models Analysis; LS mean difference = 0.49, 95% CI 2-sided [0.19 to 0.78], Standard Error of Mean 0.148
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.0008, Mixed Models Analysis; LS mean difference = 0.48, 95% CI 2-sided [0.20 to 0.76], Standard Error of Mean 0.142
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0004, Mixed Models Analysis; LS mean difference = 0.53, 95% CI 2-sided [0.24 to 0.81], Standard Error of Mean 0.147
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0918, Mixed Models Analysis; LS mean difference = 0.32, 95% CI 2-sided [-0.05 to 0.69], Standard Error of Mean 0.188
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.1600, Mixed Models Analysis; LS mean difference = 0.25, 95% CI 2-sided [-0.10 to 0.61], Standard Error of Mean 0.179
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.6776, Mixed Models Analysis; LS mean difference = 0.08, 95% CI 2-sided [-0.30 to 0.47], Standard Error of Mean 0.195
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.5646, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-0.25 to 0.46], Standard Error of Mean 0.180

19. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Scores: Tragus-to-wall Distance at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASMI assessed axial status and spinal mobility, using linear function. It composed of 5 clinical measures: lateral spinal flexion, tragus-to-wall distance, lumbar flexion (modified Schober), maximal intermalleolar distance, cervical rotation. BASMI - Linear Method score was average of 5 individual component scores mapped between 0 and 10, with higher scores indicating more impairment of axial status and spinal mobility. For the assessment of tragus-to-wall distance, participant was placed standing with his/her back against the wall; knees straight; scapulae, buttocks, and heels against wall; and head in as neutral position as possible. The distance between the tragus and wall in cm was measured (to the nearest 0.1 cm) from both the right side and left side at the maximum effort to touch the head against the wall. Distance should be greater than or equal to 0 cm with no defined maximum value, lower tragus-to-wall value indicates better health status.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Centimeters
  Week 2 | -0.19 (0.126) | -0.24 (0.125)
  Week 4 | -0.48 (0.144) | -0.07 (0.143)
  Week 8 | -0.51 (0.177) | 0.36 (0.177)
  Week 12 | -0.40 (0.169) | 0.23 (0.169)
  Week 16 | -0.50 (0.168) | 0.09 (0.168)
  Week 24 | -0.66 (0.202) | -0.03 (0.201)
  Week 32 | -0.66 (0.179) | 0.00 (0.178)
  Week 40 | -0.60 (0.200) | -0.14 (0.199)
  Week 48 | -0.73 (0.204) | -0.18 (0.202)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.7291, Mixed Models Analysis; LS mean difference = 0.06, 95% CI 2-sided [-0.26 to 0.37], Standard Error of Mean 0.161
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0257, Mixed Models Analysis; LS mean difference = -0.41, 95% CI 2-sided [-0.78 to -0.05], Standard Error of Mean 0.184
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS mean difference = -0.86, 95% CI 2-sided [-1.31 to -0.42], Standard Error of Mean 0.227
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.0041, Mixed Models Analysis; LS mean difference = -0.63, 95% CI 2-sided [-1.05 to -0.20], Standard Error of Mean 0.216
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0062, Mixed Models Analysis; LS mean difference = -0.59, 95% CI 2-sided [-1.02 to -0.17], Standard Error of Mean 0.215
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0140, Mixed Models Analysis; LS mean difference = -0.63, 95% CI 2-sided [-1.13 to -0.13], Standard Error of Mean 0.255
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0035, Mixed Models Analysis; LS mean difference = -0.66, 95% CI 2-sided [-1.11 to -0.22], Standard Error of Mean 0.225
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0645, Mixed Models Analysis; LS mean difference = -0.47, 95% CI 2-sided [-0.97 to 0.03], Standard Error of Mean 0.253
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0341, Mixed Models Analysis; LS mean difference = -0.54, 95% CI 2-sided [-1.05 to -0.04], Standard Error of Mean 0.255

20. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Linear Method Total Score at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: The BASMI was used to assess the axial status and spinal mobility (cervical, dorsal and lumbar spine, hips and pelvic soft tissue) and was analyzed using the linear function method. BASMI score composed of five clinical measures: lateral spinal flexion, tragus-to-wall distance, lumbar flexion (modified Schober), maximal intermalleolar distance, and cervical rotation. BASMI - Linear Method score was the average of 5 individual component scores mapped between 0 and 10 and thus the BASMI - Linear Method total score ranged from 0 (very good) to 10 (very poor), wherein higher scores indicated more impairment of axial status and spinal mobility; lower scores indicated better health status.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -0.25 (0.044) | -0.03 (0.043)
  Week 4 | -0.39 (0.053) | -0.06 (0.053)
  Week 8 | -0.49 (0.059) | -0.03 (0.058)
  Week 12 | -0.49 (0.058) | -0.02 (0.058)
  Week 16 | -0.63 (0.060) | -0.11 (0.060)
  Week 24 | -0.67 (0.068) | -0.38 (0.068)
  Week 32 | -0.74 (0.069) | -0.52 (0.068)
  Week 40 | -0.74 (0.074) | -0.55 (0.073)
  Week 48 | -0.69 (0.074) | -0.54 (0.073)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LS mean difference = -0.22, 95% CI 2-sided [-0.33 to -0.11], Standard Error of Mean 0.056
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.33, 95% CI 2-sided [-0.47 to -0.20], Standard Error of Mean 0.068
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.46, 95% CI 2-sided [-0.61 to -0.31], Standard Error of Mean 0.075
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.47, 95% CI 2-sided [-0.62 to -0.32], Standard Error of Mean 0.075
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.52, 95% CI 2-sided [-0.67 to -0.37], Standard Error of Mean 0.077
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0008, LS mean difference; LS mean difference = -0.29, 95% CI 2-sided [-0.46 to -0.12], Standard Error of Mean 0.086
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0116, Mixed Models Analysis; LS mean difference = -0.22, 95% CI 2-sided [-0.39 to -0.05], Standard Error of Mean 0.086
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0416, Mixed Models Analysis; LS mean difference = -0.19, 95% CI 2-sided [-0.37 to -0.01], Standard Error of Mean 0.093
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0915, Mixed Models Analysis; LS mean difference = -0.16, 95% CI 2-sided [-0.34 to 0.03], Standard Error of Mean 0.092

21. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Total Scores at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: FACIT-F is a 13-item questionnaire (felt fatigued, felt weak all over, felt listless ["washed out"],felt tired, had energy, had trouble starting things as tired, had trouble finishing things as tired, was able to do usual activities, needed to sleep during day, too tired to eat, needed help doing my usual activities, frustrated by being too tired to do things wanted to do, had to limit my social activity because tired), with each item scored on a 5-point scale ranging from 0 (not at all) to 4 (very much). Three type of scores were derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score was calculated by summing the 13 items (range 0 [not at all] to 52 [very much]); higher scores represent less fatigue status. In this outcome measure, change from baseline in FACIT-F total score was reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | 3.16 (0.552) | 0.32 (0.548)
  Week 4 | 4.80 (0.595) | 1.19 (0.591)
  Week 8 | 6.46 (0.706) | 1.03 (0.703)
  Week 12 | 6.25 (0.737) | 1.24 (0.736)
  Week 16 | 6.54 (0.795) | 3.12 (0.794)
  Week 24 | 7.42 (0.842) | 5.84 (0.836)
  Week 32 | 7.90 (0.813) | 7.24 (0.807)
  Week 40 | 8.67 (0.817) | 7.15 (0.810)
  Week 48 | 9.54 (0.897) | 7.35 (0.891)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 2.85, 95% CI 2-sided [1.46 to 4.24], Standard Error of Mean 0.706
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 3.61, 95% CI 2-sided [2.11 to 5.10], Standard Error of Mean 0.761
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 5.42, 95% CI 2-sided [3.65 to 7.20], Standard Error of Mean 0.902
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 5.01, 95% CI 2-sided [3.15 to 6.86], Standard Error of Mean 0.943
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0008, Mixed Models Analysis; LS mean difference = 3.43, 95% CI 2-sided [1.44 to 5.42], Standard Error of Mean 1.012
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.1390, Mixed Models Analysis; LS mean difference = 1.58, 95% CI 2-sided [-0.52 to 3.68], Standard Error of Mean 1.064
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.5217, Mixed Models Analysis; LS mean difference = 0.66, 95% CI 2-sided [-1.36 to 2.67], Standard Error of Mean 1.024
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.1415, Mixed Models Analysis; LS mean difference = 1.51, 95% CI 2-sided [-0.51 to 3.54], Standard Error of Mean 1.027
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0533, Mixed Models Analysis; LS mean difference = 2.19, 95% CI 2-sided [-0.03 to 4.41], Standard Error of Mean 1.128

22. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Experience Domain Scores at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: FACIT-F is a 13-item (felt fatigued, felt weak all over, felt listless ["washed out"],felt tired, had energy, had trouble starting things as tired, had trouble finishing things as tired, was able to do usual activities, needed to sleep during day, too tired to eat, needed help doing my usual activities, frustrated by being too tired to do things wanted to do, had to limit my social activity because tired) questionnaire, with each item scored on a 5-point scale ranging from 0 (not at all) to 4 (very much). FACIT-F experience domain score was calculated by summing 5 items: I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy. FACIT-F total experience domain score ranged from 0 (not at all) to 20 (very much), with higher scores represented better (less) fatigue impact on daily functioning. In this outcome measure, change from baseline in FACIT-F experience domain score was reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | 1.35 (0.275) | 0.11 (0.274)
  Week 4 | 2.30 (0.298) | 0.60 (0.296)
  Week 8 | 2.72 (0.331) | 0.53 (0.330)
  Week 12 | 2.78 (0.343) | 0.80 (0.344)
  Week 16 | 2.85 (0.357) | 1.29 (0.357)
  Week 24 | 3.58 (0.384) | 2.96 (0.382)
  Week 32 | 3.65 (0.370) | 3.43 (0.367)
  Week 40 | 3.98 (0.375) | 3.59 (0.371)
  Week 48 | 4.22 (0.403) | 3.40 (0.400)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0005, Mixed Models Analysis; LS mean difference = 1.25, 95% CI 2-sided [0.55 to 1.94], Standard Error of Mean 0.352
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 1.70, 95% CI 2-sided [0.95 to 2.45], Standard Error of Mean 0.381
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 2.19, 95% CI 2-sided [1.35 to 3.02], Standard Error of Mean 0.423
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 1.98, 95% CI 2-sided [1.11 to 2.84], Standard Error of Mean 0.439
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0007, Mixed Models Analysis; LS mean difference = 1.56, 95% CI 2-sided [0.67 to 2.45], Standard Error of Mean 0.454
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.2018, Mixed Models Analysis; LS mean difference = 0.62, 95% CI 2-sided [-0.33 to 1.58], Standard Error of Mean 0.485
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.6432, Mixed Models Analysis; LS mean difference = 0.22, 95% CI 2-sided [-0.70 to 1.13], Standard Error of Mean 0.465
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.4092, Mixed Models Analysis; LS mean difference = 0.39, 95% CI 2-sided [-0.54 to 1.31], Standard Error of Mean 0.470
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.1070, Mixed Models Analysis; LS mean difference = 0.82, 95% CI 2-sided [-0.18 to 1.81], Standard Error of Mean 0.506

23. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Impact Domain Scores at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: FACIT-F is a 13-item (felt fatigued, felt weak all over, felt listless ["washed out"],felt tired, had energy, had trouble starting things as tired, had trouble finishing things as tired, was able to do usual activities, needed to sleep during day, too tired to eat, needed help doing my usual activities, frustrated by being too tired to do things wanted to do, had to limit my social activity because tired) questionnaire, with each item scored on a 5-point scale ranging from 0 (not at all) to 4 (very much). FACIT-F experience domain score calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless, I feel tired, and I have energy, while FACIT-F impact domain score was calculated by summing the remaining 8 items. FACIT-F impact domain score ranged from 0 (not at all) to 32 (very much), with higher scores represented better (less) fatigue impact on daily functioning. In this outcome measure, change from baseline in FACIT-F impact domain score was reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | 1.79 (0.334) | 0.17 (0.332)
  Week 4 | 2.47 (0.364) | 0.55 (0.361)
  Week 8 | 3.73 (0.429) | 0.46 (0.428)
  Week 12 | 3.45 (0.440) | 0.41 (0.441)
  Week 16 | 3.68 (0.488) | 1.81 (0.487)
  Week 24 | 3.84 (0.504) | 2.86 (0.501)
  Week 32 | 4.25 (0.489) | 3.80 (0.485)
  Week 40 | 4.70 (0.480) | 3.57 (0.476)
  Week 48 | 5.32 (0.542) | 3.95 (0.538)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS mean difference = 1.62, 95% CI 2-sided [0.78 to 2.46], Standard Error of Mean 0.428
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 1.92, 95% CI 2-sided [1.00 to 2.84], Standard Error of Mean 0.466
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 3.26, 95% CI 2-sided [2.18 to 4.34], Standard Error of Mean 0.549
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = 3.04, 95% CI 2-sided [1.93 to 4.15], Standard Error of Mean 0.564
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0028, Mixed Models Analysis; LS mean difference = 1.87, 95% CI 2-sided [0.65 to 3.09], Standard Error of Mean 0.621
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.1289, Mixed Models Analysis; LS mean difference = 0.97, 95% CI 2-sided [-0.28 to 2.23], Standard Error of Mean 0.638
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.4698, Mixed Models Analysis; LS mean difference = 0.45, 95% CI 2-sided [-0.77 to 1.66], Standard Error of Mean 0.616
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0616, Mixed Models Analysis; LS mean difference = 1.13, 95% CI 2-sided [-0.06 to 2.32], Standard Error of Mean 0.603
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0455, Mixed Models Analysis; LS mean difference = 1.37, 95% CI 2-sided [0.03 to 2.71], Standard Error of Mean 0.681

24. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease (PGA) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Participants answered the question, "How active was your spondylitis on average during the last week?. Participant's response was recorded using a numerical rating scale ranged from 0 (Not Active) to 10 (Very Active), with higher scores indicated more severe disease.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -1.21 (0.144) | -0.32 (0.144)
  Week 4 | -1.85 (0.168) | -0.63 (0.167)
  Week 8 | -2.14 (0.181) | -0.42 (0.181)
  Week 12 | -2.37 (0.193) | -0.65 (0.193)
  Week 16 | -2.47 (0.204) | -0.91 (0.204)
  Week 24 | -2.76 (0.222) | -2.21 (0.221)
  Week 32 | -3.04 (0.228) | -2.43 (0.226)
  Week 40 | -3.04 (0.222) | -2.50 (0.220)
  Week 48 | -3.47 (0.225) | -2.94 (0.223)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.88, 95% CI 2-sided [-1.25 to -0.52], Standard Error of Mean 0.185
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.22, 95% CI 2-sided [-1.65 to -0.80], Standard Error of Mean 0.215
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.71, 95% CI 2-sided [-2.17 to -1.26], Standard Error of Mean 0.232
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.72, 95% CI 2-sided [-2.20 to -1.23], Standard Error of Mean 0.247
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.56, 95% CI 2-sided [-2.07 to -1.05], Standard Error of Mean 0.260
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0483, Mixed Models Analysis; LS mean difference = -0.56, 95% CI 2-sided [-1.11 to -0.00], Standard Error of Mean 0.281
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0357, Mixed Models Analysis; LS mean difference = -0.60, 95% CI 2-sided [-1.17 to -0.04], Standard Error of Mean 0.286
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0508, Mixed Models Analysis; LS mean difference = -0.55, 95% CI 2-sided [-1.09 to 0.00], Standard Error of Mean 0.278
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0614, Mixed Models Analysis; LS mean difference = -0.53, 95% CI 2-sided [-1.08 to 0.03], Standard Error of Mean 0.282

25. Secondary Outcome: Change From Baseline in Patient's Assessment of Spinal Pain: Total Back Pain at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Participants marked their level of total back pain on a numerical rating scale (NRS) ranged from 0 (no pain) to 10 (most severe pain), with higher scores indicated more severe pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -1.28 (0.145) | -0.38 (0.144)
  Week 4 | -2.05 (0.164) | -0.71 (0.164)
  Week 8 | -2.51 (0.173) | -0.53 (0.173)
  Week 12 | -2.57 (0.192) | -0.69 (0.192)
  Week 16 | -2.57 (0.191) | -0.96 (0.191)
  Week 24 | -2.99 (0.206) | -2.47 (0.205)
  Week 32 | -3.16 (0.212) | -2.86 (0.210)
  Week 40 | -3.11 (0.217) | -2.62 (0.215)
  Week 48 | -3.57 (0.220) | -2.87 (0.218)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.89, 95% CI 2-sided [-1.26 to -0.53], Standard Error of Mean 0.186
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.34, 95% CI 2-sided [-1.75 to -0.92], Standard Error of Mean 0.210
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.98, 95% CI 2-sided [-2.41 to -1.54], Standard Error of Mean 0.221
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.89, 95% CI 2-sided [-2.37 to -1.40], Standard Error of Mean 0.245
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.62, 95% CI 2-sided [-2.10 to -1.14], Standard Error of Mean 0.243
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0492, Mixed Models Analysis; LS mean difference = -0.51, 95% CI 2-sided [-1.03 to -0.00], Standard Error of Mean 0.261
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.2614, Mixed Models Analysis; LS mean difference = -0.30, 95% CI 2-sided [-0.82 to 0.22], Standard Error of Mean 0.266
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0722, Mixed Models Analysis; LS mean difference = -0.49, 95% CI 2-sided [-1.03 to 0.04], Standard Error of Mean 0.272
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0121, Mixed Models Analysis; LS mean difference = -0.70, 95% CI 2-sided [-1.24 to -0.15], Standard Error of Mean 0.275

26. Secondary Outcome: Change From Baseline in Patient's Assessment of Spinal Pain: Nocturnal Spinal Pain at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Participants marked their level of nocturnal spinal pain on a NRS ranged from 0 (no pain) to 10 (most severe pain), with higher scores indicated more severe pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -1.24 (0.162) | -0.32 (0.161)
  Week 4 | -2.15 (0.169) | -0.56 (0.167)
  Week 8 | -2.61 (0.191) | -0.59 (0.190)
  Week 12 | -2.60 (0.198) | -0.60 (0.199)
  Week 16 | -2.67 (0.204) | -0.84 (0.204)
  Week 24 | -3.07 (0.217) | -2.59 (0.215)
  Week 32 | -3.17 (0.219) | -2.89 (0.217)
  Week 40 | -3.20 (0.226) | -2.73 (0.224)
  Week 48 | -3.52 (0.229) | -3.01 (0.227)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.92, 95% CI 2-sided [-1.33 to -0.51], Standard Error of Mean 0.207
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.60, 95% CI 2-sided [-2.02 to -1.17], Standard Error of Mean 0.216
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -2.02, 95% CI 2-sided [-2.50 to -1.54], Standard Error of Mean 0.244
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -2.00, 95% CI 2-sided [-2.50 to -1.50], Standard Error of Mean 0.254
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.84, 95% CI 2-sided [-2.35 to -1.32], Standard Error of Mean 0.260
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0785, Mixed Models Analysis; LS mean difference = -0.48, 95% CI 2-sided [-1.02 to 0.06], Standard Error of Mean 0.274
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.3047, Mixed Models Analysis; LS mean difference = -0.28, 95% CI 2-sided [-0.82 to 0.26], Standard Error of Mean 0.275
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.1009, Mixed Models Analysis; LS mean difference = -0.47, 95% CI 2-sided [-1.02 to 0.09], Standard Error of Mean 0.283
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0764, Mixed Models Analysis; LS mean difference = -0.51, 95% CI 2-sided [-1.08 to 0.05], Standard Error of Mean 0.287

27. Secondary Outcome: Change From Baseline in in Bath Ankylosing Spondylitis Functional Index (BASFI) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASFI was a functional index which included 10 items assessing ability of participants to perform normal daily activities. The first 8 questions/items consider activities related to functional anatomy. The final 2 questions/items assess the participants' ability to cope with everyday life. Each item was scored on a scale of 0=easy to 10=impossible. The BASFI total score was calculated as the average score of these 10 individual items. BASFI total score ranged from 0 (easy) to 10 (impossible), where higher scores indicated more severe disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -0.87 (0.125) | -0.45 (0.124)
  Week 4 | -1.35 (0.140) | -0.58 (0.139)
  Week 8 | -1.79 (0.158) | -0.69 (0.157)
  Week 12 | -2.01 (0.164) | -0.71 (0.164)
  Week 16 | -2.05 (0.170) | -0.82 (0.169)
  Week 24 | -2.25 (0.191) | -1.91 (0.190)
  Week 32 | -2.42 (0.188) | -2.16 (0.187)
  Week 40 | -2.62 (0.192) | -2.23 (0.191)
  Week 48 | -2.61 (0.196) | -2.32 (0.195)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0089, Mixed Models Analysis; LS mean difference = -0.42, 95% CI 2-sided [-0.73 to -0.11], Standard Error of Mean 0.159
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.77, 95% CI 2-sided [-1.12 to -0.42], Standard Error of Mean 0.179
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.10, 95% CI 2-sided [-1.50 to -0.70], Standard Error of Mean 0.202
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.29, 95% CI 2-sided [-1.71 to -0.88], Standard Error of Mean 0.210
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.23, 95% CI 2-sided [-1.66 to -0.80], Standard Error of Mean 0.217
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.1686, Mixed Models Analysis; LS mean difference = -0.33, 95% CI 2-sided [-0.81 to 0.14], Standard Error of Mean 0.242
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.2800, Mixed Models Analysis; LS mean difference = -0.26, 95% CI 2-sided [-0.72 to 0.21], Standard Error of Mean 0.238
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.1135, Mixed Models Analysis; LS mean difference = -0.39, 95% CI 2-sided [-0.86 to 0.09], Standard Error of Mean 0.243
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.2496, Mixed Models Analysis; LS mean difference = -0.29, 95% CI 2-sided [-0.77 to 0.20], Standard Error of Mean 0.247

28. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Inflammation (Morning Stiffness) Score at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: The BASDAI was a validated questionnaire that consisted of 6 questions pertaining to the 5 major symptoms of AS: fatigue; spinal pain; peripheral arthritis; enthesitis, intensity of morning stiffness and duration of morning stiffness. Each question was rated using a numerical rating scale from 0 (none) to 10 (very severe), higher score=high disease activity. The BASDAI score was calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions 1 to 4. This score was then divided by 5. The total BASDAI score was ranged from 0= none to 10= very severe, where higher score indicated high disease activity. BASDAI inflammation score was derived by taking mean of the responses of question 5 and 6 and ranged from 0 (none) to 10 (very severe), where higher score indicated more inflammation (morning stiffness).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -1.33 (0.149) | -0.49 (0.149)
  Week 4 | -2.08 (0.164) | -0.60 (0.163)
  Week 8 | -2.52 (0.178) | -0.91 (0.178)
  Week 12 | -2.71 (0.185) | -0.84 (0.186)
  Week 16 | -2.69 (0.185) | -0.97 (0.185)
  Week 24 | -2.99 (0.193) | -2.48 (0.193)
  Week 32 | -3.11 (0.200) | -2.61 (0.199)
  Week 40 | -3.28 (0.204) | -2.64 (0.203)
  Week 48 | -3.46 (0.214) | -2.90 (0.213)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.84, 95% CI 2-sided [-1.22 to -0.47], Standard Error of Mean 0.191
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.48, 95% CI 2-sided [-1.89 to -1.07], Standard Error of Mean 0.210
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.61, 95% CI 2-sided [-2.06 to -1.16], Standard Error of Mean 0.228
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.87, 95% CI 2-sided [-2.34 to -1.40], Standard Error of Mean 0.237
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.72, 95% CI 2-sided [-2.18 to -1.25], Standard Error of Mean 0.236
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0385, Mixed Models Analysis; LS mean difference = -0.51, 95% CI 2-sided [-0.99 to -0.03], Standard Error of Mean 0.245
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0463, Mixed Models Analysis; LS mean difference = -0.50, 95% CI 2-sided [-1.00 to -0.01], Standard Error of Mean 0.252
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0126, Mixed Models Analysis; LS mean difference = -0.65, 95% CI 2-sided [-1.15 to -0.14], Standard Error of Mean 0.257
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0372, Mixed Models Analysis; LS mean difference = -0.56, 95% CI 2-sided [-1.09 to -0.03], Standard Error of Mean 0.268

29. Secondary Outcome: Percentage of Participants Achieving ASAS 5/6 Response at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: ASAS 5/6 consists of 6 domains: 4 used in ASAS20 - PGA (assess disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity), Spinal Pain (total back pain) (on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity), Function (using BASFI which assess participant's level of ability on a scale of 0 [easy] to 10 [impossible], lower scores= better functional health) and Inflammation (using BASDAI, mean of Q 5 and 6, which assess disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity), CRP (was measured in mg per liter) and Spinal mobility was measured in centimeter and calculated as mean of right and left measurements of lateral spinal flexion from BASMI. ASAS 5/6: defined as >=20% improvement in at least 5 domains.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants
  Week 2 | 16.54 | 2.94
  Week 4 | 35.34 | 6.62
  Week 8 | 41.35 | 8.09
  Week 12 | 45.86 | 9.56
  Week 16 | 43.61 | 7.35
  Week 24 | 49.62 | 44.12
  Week 32 | 51.13 | 53.68
  Week 40 | 48.87 | 50.74
  Week 48 | 43.61 | 44.85
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 13.60, 95% CI 2-sided [6.68 to 20.52], Standard Error of Mean 3.53
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 28.79, 95% CI 2-sided [19.78 to 37.80], Standard Error of Mean 4.60
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 33.31, 95% CI 2-sided [23.84 to 42.78], Standard Error of Mean 4.83
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 36.37, 95% CI 2-sided [26.67 to 46.07], Standard Error of Mean 4.95
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16: Analysis performed using Normal approximation adjusting for the stratification factor derived from clinical database via CMH approach; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 36.34, 95% CI 2-sided [27.05 to 45.63], Standard Error of Mean 4.74
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.3498, Cochran-Mantel-Haenszel; Difference in percentage = 5.60, 95% CI 2-sided [-6.14 to 17.35], Standard Error of Mean 5.99
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.6835, Cochran-Mantel-Haenszel; Difference in percentage = -2.40, 95% CI 2-sided [-13.96 to 9.15], Standard Error of Mean 5.89
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.7704, Cochran-Mantel-Haenszel; Difference in percentage = -1.75, 95% CI 2-sided [-13.47 to 9.98], Standard Error of Mean 5.98
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.8492, Cochran-Mantel-Haenszel; Difference in percentage = -1.13, 95% CI 2-sided [-12.80 to 10.53], Standard Error of Mean 5.95

30. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Partial remission was defined as a score of 2 or less (on a scale of 0-10, where 0=no disease activity and 10=high disease activity) in each of the 4 domains in ASAS. These 4 domains included: PGA (assess disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity), total back pain (on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity), Function (using BASFI which assess participant's level of ability on a scale of 0 [easy] to 10 [impossible], lower scores= better functional health) and Inflammation (using BASDAI, mean of Q 5 and 6, which assess disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity).
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants
  Week 2 | 2.26 | 0
  Week 4 | 4.51 | 0
  Week 8 | 7.52 | 1.47
  Week 12 | 15.04 | 2.94
  Week 16 | 15.04 | 2.94
  Week 24 | 21.80 | 11.76
  Week 32 | 23.31 | 15.44
  Week 40 | 24.06 | 16.91
  Week 48 | 23.31 | 17.65
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.1692, Cochran-Mantel-Haenszel; Difference in percentage = 2.24, 95% CI 2-sided [-0.95 to 5.43], Standard Error of Mean 1.63
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.0289, Cochran-Mantel-Haenszel; Difference in percentage = 4.46, 95% CI 2-sided [0.46 to 8.46], Standard Error of Mean 2.04
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.0199, Cochran-Mantel-Haenszel; Difference in percentage = 6.02, 95% CI 2-sided [0.95 to 11.09], Standard Error of Mean 2.59
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.0005, Difference in percentage; Difference in percentage = 12.03, 95% CI 2-sided [5.26 to 18.81], Standard Error of Mean 3.46
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 29, analysis 5]; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Difference in percentage = 12.05, 95% CI 2-sided [5.29 to 18.80], Standard Error of Mean 3.45
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.0253, Cochran-Mantel-Haenszel; Difference in percentage = 10.03, 95% CI 2-sided [1.24 to 18.83], Standard Error of Mean 4.49
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.0950, Cochran-Mantel-Haenszel; Difference in percentage = 7.93, 95% CI 2-sided [-1.38 to 17.24], Standard Error of Mean 4.75
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.1377, Cochran-Mantel-Haenszel; Difference in percentage = 7.21, 95% CI 2-sided [-2.31 to 16.73], Standard Error of Mean 4.86
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.2472, Cochran-Mantel-Haenszel; Difference in percentage = 5.68, 95% CI 2-sided [-3.94 to 15.30], Standard Error of Mean 4.91

31. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: The BASDAI was a validated questionnaire that consisted of 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: fatigue; spinal pain; peripheral arthritis; enthesitis, intensity of morning stiffness and duration of morning stiffness. Each question was rated using a numerical rating scale from 0 (none) to 10 (very severe), higher score=high disease activity. The BASDAI score was calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions 1 to 4. This score was then divided by 5. The total BASDAI score was ranged from 0= none to 10= very severe, where higher score indicated high disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Units on a scale
  Week 2 | -1.25 (0.127) | -0.52 (0.126)
  Week 4 | -1.95 (0.146) | -0.67 (0.145)
  Week 8 | -2.32 (0.164) | -0.82 (0.163)
  Week 12 | -2.49 (0.172) | -0.81 (0.172)
  Week 16 | -2.55 (0.175) | -1.11 (0.174)
  Week 24 | -2.81 (0.185) | -2.41 (0.184)
  Week 32 | -2.94 (0.191) | -2.53 (0.190)
  Week 40 | -3.09 (0.193) | -2.63 (0.192)
  Week 48 | -3.30 (0.199) | -2.80 (0.197)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -0.73, 95% CI 2-sided [-1.05 to -0.41], Standard Error of Mean 0.163
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.28, 95% CI 2-sided [-1.65 to -0.91], Standard Error of Mean 0.187
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.50, 95% CI 2-sided [-1.92 to -1.09], Standard Error of Mean 0.210
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.68, 95% CI 2-sided [-2.11 to -1.24], Standard Error of Mean 0.221
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.44, 95% CI 2-sided [-1.88 to -1.00], Standard Error of Mean 0.223
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0880, Mixed Models Analysis; LS mean difference = -0.40, 95% CI 2-sided [-0.86 to 0.06], Standard Error of Mean 0.235
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0921, Mixed Models Analysis; LS mean difference = -0.41, 95% CI 2-sided [-0.88 to 0.07], Standard Error of Mean 0.241
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.0597, Mixed Models Analysis; LS mean difference = -0.46, 95% CI 2-sided [-0.94 to 0.02], Standard Error of Mean 0.243
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0492, Mixed Models Analysis; LS mean difference = -0.49, 95% CI 2-sided [-0.99 to -0.00], Standard Error of Mean 0.250

32. Secondary Outcome: Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI50) Response at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: BASDAI was a validated questionnaire that consisted of 6 questions pertaining to the 5 major symptoms of AS: fatigue; spinal pain; peripheral arthritis; enthesitis, intensity of morning stiffness and duration of morning stiffness. Each question was rated using a numerical rating scale from 0 (none) to 10 (very severe), higher score=high disease activity. BASDAI score was calculated by computing mean of questions 5 and 6 and adding it to sum of questions 1 to 4. This score was then divided by 5. The total BASDAI score was ranged from 0= none to 10= very severe, where higher score indicated high disease activity. BASDAI50 response was defined as decrease of >=50% from Baseline in BASDAI score at specified time points. Percentage of participants with BASDAI 50 response at specified weeks are reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants
  Week 2 | 12.03 | 3.68
  Week 4 | 29.32 | 6.62
  Week 8 | 39.85 | 11.03
  Week 12 | 42.86 | 11.03
  Week 16 | 42.86 | 17.65
  Week 24 | 47.37 | 36.76
  Week 32 | 51.13 | 41.18
  Week 40 | 52.63 | 39.71
  Week 48 | 51.13 | 40.44
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0116, Cochran-Mantel-Haenszel; Difference in percentage = 8.31, 95% CI 2-sided [1.86 to 14.77], Standard Error of Mean 3.29
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 22.74, 95% CI 2-sided [13.99 to 31.49], Standard Error of Mean 4.46
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 28.87, 95% CI 2-sided [19.09 to 38.66], Standard Error of Mean 4.99
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 31.93, 95% CI 2-sided [22.28 to 41.58], Standard Error of Mean 4.92
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 29, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 25.28, 95% CI 2-sided [14.82 to 35.75], Standard Error of Mean 5.34
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.0683, Cochran-Mantel-Haenszel; Difference in percentage = 10.71, 95% CI 2-sided [-0.80 to 22.23], Standard Error of Mean 5.88
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.0906, Cochran-Mantel-Haenszel; Difference in percentage = 10.05, 95% CI 2-sided [-1.59 to 21.70], Standard Error of Mean 5.94
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.0282, Cochran-Mantel-Haenszel; Difference in percentage = 13.03, 95% CI 2-sided [1.39 to 24.66], Standard Error of Mean 5.94
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.0719, Cochran-Mantel-Haenszel; Difference in percentage = 10.77, 95% CI 2-sided [-0.96 to 22.49], Standard Error of Mean 5.98

33. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score Using C-Reactive Protein (ASDAS[CRP]) Clinically Important Improvement Response at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: ASDAS(CRP) was derived using BASDAI (6-item questionnaire measures disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and PGA (measure disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity) and by using the following formula, 0.121 x Back Pain (Q2 of BASDAI) + 0.058 x Duration of Morning Stiffness (Q6 of BASDAI) + 0.110 x PGA + 0.073 x Peripheral Pain/Swelling (Q3 of BASDAI) + 0.579 x Ln(hsCRP mg/L + 1). If hsCRP values were smaller than 2 mg/L, they were set to 2 mg/L in the formula. The range of score was >= 0.636 to no defined upper limit. A negative change from baseline value indicates decrease in disease activity; a positive change from baseline value indicates increase in disease activity. ASDAS(CRP) clinically important improvement was defined as decrease from Baseline of >=1.1 units in ASDAS(CRP) score.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Analysis included only participants with baseline ASDAS(CRP) >= 1.736 units. Here, on-drug data was used and missing response (MR) was considered to be Non-response (NR) (MR=NR). Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Percentage of participants
  Week 2 | 39.39 | 6.62
  Week 4 | 53.03 | 12.50
  Week 8 | 59.85 | 14.71
  Week 12 | 60.61 | 15.44
  Week 16 | 61.36 | 19.12
  Week 24 | 65.15 | 60.29
  Week 32 | 65.91 | 61.76
  Week 40 | 63.64 | 57.35
  Week 48 | 58.33 | 52.94
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 32.79, 95% CI 2-sided [23.48 to 42.11], Standard Error of Mean 4.75
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 40.53, 95% CI 2-sided [30.37 to 50.70], Standard Error of Mean 5.19
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 45.22, 95% CI 2-sided [35.03 to 55.41], Standard Error of Mean 5.20
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 45.23, 95% CI 2-sided [34.97 to 55.49], Standard Error of Mean 5.23
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 29, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 42.30, 95% CI 2-sided [31.73 to 52.88], Standard Error of Mean 5.40
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.3967, Cochran-Mantel-Haenszel; Difference in percentage = 4.96, 95% CI 2-sided [-6.51 to 16.42], Standard Error of Mean 5.85
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.4442, Cochran-Mantel-Haenszel; Difference in percentage = 4.34, 95% CI 2-sided [-6.78 to 15.46], Standard Error of Mean 5.67
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.2810, Cochran-Mantel-Haenszel; Difference in percentage = 6.38, 95% CI 2-sided [-5.22 to 17.97], Standard Error of Mean 5.92
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.3514, Cochran-Mantel-Haenszel; Difference in percentage = 5.54, 95% CI 2-sided [-6.12 to 17.20], Standard Error of Mean 5.95

34. Secondary Outcome: Percentage of Participants Ankylosing Spondylitis Disease Activity Score Using C-Reactive Protein (ASDAS[CRP]) Major Improvement Response at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: ASDAS(CRP) was derived using BASDAI (6-item questionnaire measures disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and PGA (measure disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity) and by using the following formula, 0.121 x Back Pain (Q2 of BASDAI) + 0.058 x Duration of Morning Stiffness (Q6 of BASDAI) + 0.110 x PGA + 0.073 x Peripheral Pain/Swelling (Q3 of BASDAI) + 0.579 x Ln(hsCRP mg/L + 1). If hsCRP values were smaller than 2 mg/L, they were set to 2 mg/L in the formula. The range of score was >= 0.636 to no defined upper limit. A negative change from baseline value indicates decrease in disease activity; a positive change from baseline value indicates increase in disease activity. ASDAS(CRP) major improvement was defined as a response if improvement (decrease) from Baseline in ASDAS(CRP) of >=2.0 units.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Analysis included only participants with baseline ASDAS(CRP) >= 2.636 units. Here, on-drug data was used and missing response (MR) was considered to be Non-response (NR) (MR=NR). Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 123 | 129
Percentage of participants
  Week 2 | 8.94 | 0.00
  Week 4 | 17.89 | 1.55
  Week 8 | 22.76 | 2.33
  Week 12 | 26.02 | 3.10
  Week 16 | 30.08 | 4.65
  Week 24 | 34.15 | 24.81
  Week 32 | 36.59 | 34.11
  Week 40 | 39.02 | 31.78
  Week 48 | 33.33 | 28.68
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Difference in percentage = 8.84, 95% CI 2-sided [3.46 to 14.21], Standard Error of Mean 2.74
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 16.25, 95% CI 2-sided [9.13 to 23.36], Standard Error of Mean 3.63
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 20.31, 95% CI 2-sided [12.41 to 28.20], Standard Error of Mean 4.03
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 22.77, 95% CI 2-sided [14.46 to 31.08], Standard Error of Mean 4.24
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 29, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 25.28, 95% CI 2-sided [16.47 to 34.10], Standard Error of Mean 4.50
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.0941, Cochran-Mantel-Haenszel; Difference in percentage = 9.41, 95% CI 2-sided [-1.61 to 20.43], Standard Error of Mean 5.62
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.6727, Cochran-Mantel-Haenszel; Difference in percentage = 2.52, 95% CI 2-sided [-9.17 to 14.21], Standard Error of Mean 5.96
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.2213, Cochran-Mantel-Haenszel; Difference in percentage = 7.29, 95% CI 2-sided [-4.39 to 18.98], Standard Error of Mean 5.96
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.4137, Cochran-Mantel-Haenszel; Difference in percentage = 4.70, 95% CI 2-sided [-6.58 to 15.98], Standard Error of Mean 5.76

35. Secondary Outcome: Percentage of Participants Ankylosing Spondylitis Disease Activity Score Using C-Reactive Protein (ASDAS[CRP]) Inactive Disease Response at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: ASDAS(CRP) was derived using BASDAI (6-item questionnaire measures disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and PGA (measure disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity) and by using the following formula, 0.121 x Back Pain (Q2 of BASDAI) + 0.058 x Duration of Morning Stiffness (Q6 of BASDAI) + 0.110 x PGA + 0.073 x Peripheral Pain/Swelling (Q3 of BASDAI) + 0.579 x Ln(hsCRP mg/L + 1). If hsCRP values were smaller than 2 mg/L, they were set to 2 mg/L in the formula. The range of score was >= 0.636 to no defined upper limit. A negative change from baseline value indicates decrease in disease activity; a positive change from baseline value indicates increase in disease activity. ASDAS(CRP) inactive disease is defined as a response if actual ASDAS(CRP) was <1.3 units.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Analysis included only participants with baseline ASDAS(CRP) >= 1.3 units. Here, on-drug data was used and missing response (MR) was considered to be Non-response (NR) (MR=NR).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 133 | 136
Percentage of participants
  Week 2 | 0.75 | 0.00
  Week 4 | 3.76 | 0.00
  Week 8 | 6.02 | 0.74
  Week 12 | 11.28 | 0.74
  Week 16 | 6.77 | 0.00
  Week 24 | 12.78 | 11.76
  Week 32 | 18.05 | 13.24
  Week 40 | 17.29 | 16.91
  Week 48 | 15.04 | 13.24
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.5518, Cochran-Mantel-Haenszel; Difference in percentage = 0.75, 95% CI 2-sided [-1.73 to 3.24], Standard Error of Mean 1.27
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.0524, Cochran-Mantel-Haenszel; Difference in percentage = 3.72, 95% CI 2-sided [-0.04 to 7.47], Standard Error of Mean 1.92
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.0216, Cochran-Mantel-Haenszel; Difference in percentage = 5.25, 95% CI 2-sided [0.77 to 9.73], Standard Error of Mean 2.29
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Difference in percentage = 10.48, 95% CI 2-sided [4.80 to 16.17], Standard Error of Mean 2.90
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 29, analysis 5]; Test type: Superiority; p = 0.0047, Cochran-Mantel-Haenszel; Difference in percentage = 6.69, 95% CI 2-sided [2.05 to 11.33], Standard Error of Mean 2.37
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.7883, Cochran-Mantel-Haenszel; Difference in percentage = 1.07, 95% CI 2-sided [-6.74 to 8.88], Standard Error of Mean 3.98
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 6]; Test type: Superiority; p = 0.2708, Cochran-Mantel-Haenszel; Difference in percentage = 4.85, 95% CI 2-sided [-3.78 to 13.48], Standard Error of Mean 4.40
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 7]; Test type: Superiority; p = 0.9226, Cochran-Mantel-Haenszel; Difference in percentage = 0.44, 95% CI 2-sided [-8.48 to 9.36], Standard Error of Mean 4.55
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 9, analysis 8]; Test type: Superiority; p = 0.6630, Cochran-Mantel-Haenszel; Difference in percentage = 1.84, 95% CI 2-sided [-6.44 to 10.13], Standard Error of Mean 4.23

36. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Weeks 4, 8, 12, 16, 24, 32, 40 and 48
Description: The MASES is an index used to measure the severity of enthesitis. Enthesitis is the inflammation of enthuses (heels). The MASES assesses 13 sites for enthesitis. Sites assessed included 1st costochondral joint (left [l]/right [r]), 7th costochondral joint (l/r), posterior superior iliac spine (l/r), posterior anterior iliac spine (l/r), iliac crest (l/r), proximal insertion of Achilles tendon (l/r) and 5th lumbar spinous process. Each site was graded for the presence (1) and absence (0) of tenderness yielding total MASES score ranging from 0 (no tenderness) to 13 (worst possible score) with higher score indicated more severe tenderness.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 24, 32, 40 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Analysis included only participants with baseline MASES > 0. Here, on-drug data was used and missing response was not imputed. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 70 | 79
Units on a scale
  Week 4 | -1.42 (0.264) | -0.59 (0.244)
  Week 8 | -2.02 (0.275) | -1.28 (0.255)
  Week 12 | -1.89 (0.289) | -1.17 (0.271)
  Week 16 | -1.94 (0.288) | -1.41 (0.272)
  Week 24 | -2.50 (0.251) | -2.32 (0.240)
  Week 32 | -2.73 (0.204) | -2.54 (0.200)
  Week 40 | -2.73 (0.189) | -2.75 (0.183)
  Week 48 | -2.87 (0.225) | -2.56 (0.222)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0099, Mixed Models Analysis; LS mean difference = -0.84, 95% CI 2-sided [-1.47 to -0.20], Standard Error of Mean 0.319
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0275, Mixed Models Analysis; LS mean difference = -0.74, 95% CI 2-sided [-1.40 to -0.08], Standard Error of Mean 0.332
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.0420, Mixed Models Analysis; LS mean difference = -0.72, 95% CI 2-sided [-1.41 to -0.03], Standard Error of Mean 0.350
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.1309, Mixed Models Analysis; LS mean difference = -0.53, 95% CI 2-sided [-1.22 to 0.16], Standard Error of Mean 0.349
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.5566, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-0.78 to 0.42], Standard Error of Mean 0.305
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.4497, Mixed Models Analysis; LS mean difference = -0.19, 95% CI 2-sided [-0.68 to 0.30], Standard Error of Mean 0.248
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.9272, Mixed Models Analysis; LS mean difference = 0.02, 95% CI 2-sided [-0.43 to 0.47], Standard Error of Mean 0.227
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.2539, Mixed Models Analysis; LS mean difference = -0.31, 95% CI 2-sided [-0.85 to 0.23], Standard Error of Mean 0.273

37. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Swollen joint count was an assessment on 44 joints (sternoclaviculars, acromioclaviculars, shoulders, elbows, wrists, metacarpophalangeals, thumb interphalangeal, proximal interphalangeals, knees, ankles, and metatarsophalangeals). Each joint was assessed for swelling as: Present or Absent. Artificial joints were not assessed
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Analysis included only participants with baseline SJC(44) > 0. Here, on-drug data was used and missing response was not imputed. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Joint count
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 33 | 38
Joint count
  Week 2 | -1.71 (0.376) | -2.09 (0.358)
  Week 4 | -1.90 (0.418) | -2.23 (0.398)
  Week 8 | -2.39 (0.456) | -2.45 (0.438)
  Week 12 | -2.79 (0.428) | -2.45 (0.419)
  Week 16 | -3.35 (0.475) | -2.79 (0.465)
  Week 24 | -2.81 (0.346) | -3.32 (0.335)
  Week 32 | -2.45 (0.357) | -3.21 (0.341)
  Week 40 | -3.04 (0.289) | -3.34 (0.274)
  Week 48 | -3.31 (0.176) | -3.82 (0.174)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.4379, Mixed Models Analysis; LS mean difference = 0.37, 95% CI 2-sided [-0.58 to 1.33], Standard Error of Mean 0.479
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.5340, Mixed Models Analysis; LS mean difference = 0.33, 95% CI 2-sided [-0.73 to 1.39], Standard Error of Mean 0.532
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.9148, Mixed Models Analysis; LS mean difference = 0.06, 95% CI 2-sided [-1.10 to 1.22], Standard Error of Mean 0.582
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.5409, Mixed Models Analysis; LS mean difference = -0.34, 95% CI 2-sided [-1.43 to 0.76], Standard Error of Mean 0.548
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.3555, Mixed Models Analysis; LS mean difference = -0.57, 95% CI 2-sided [-1.78 to 0.65], Standard Error of Mean 0.607
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.2485, Mixed Models Analysis; LS mean difference = 0.51, 95% CI 2-sided [-0.36 to 1.38], Standard Error of Mean 0.436
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.0866, Mixed Models Analysis; LS mean difference = 0.76, 95% CI 2-sided [-0.11 to 1.63], Standard Error of Mean 0.435
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.4101, Mixed Models Analysis; LS mean difference = 0.30, 95% CI 2-sided [-0.42 to 1.01], Standard Error of Mean 0.356
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0237, Mixed Models Analysis; LS mean difference = 0.50, 95% CI 2-sided [0.07 to 0.94], Standard Error of Mean 0.217

38. Secondary Outcome: Change From Baseline in Spinal Mobility (Chest Expansion ) at Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Description: Chest expansion (measured in centimeters (cm), is defined as the difference in the thoracic circumference during full expiration versus full inspiration. This was measured at the 4th intercostal space. The difference between maximal inspiration and expiration of the two attempts was recorded. The better of the two attempts was used to calculate chest expansion which was defined to be greater than or equal to 0 cm with no defined maximum/upper limit. Greater chest circumference corresponds to higher score indicated more spinal mobility/better health status (measured as Chest Expansion in cm).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Centimeter
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 132 | 136
Centimeter
  Week 2 | 0.22 (0.084) | -0.09 (0.083)
  Week 4 | 0.25 (0.094) | -0.07 (0.094)
  Week 8 | 0.46 (0.114) | 0.22 (0.114)
  Week 12 | 0.57 (0.102) | 0.25 (0.102)
  Week 16 | 0.59 (0.128) | 0.38 (0.127)
  Week 24 | 0.62 (0.133) | 0.63 (0.132)
  Week 32 | 0.61 (0.149) | 0.71 (0.148)
  Week 40 | 0.75 (0.132) | 0.68 (0.131)
  Week 48 | 0.50 (0.127) | 0.47 (0.125)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0043, Mixed Models Analysis; LS mean difference = 0.31, 95% CI 2-sided [0.10 to 0.52], Standard Error of Mean 0.107
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.0072, Mixed Models Analysis; LS mean difference = 0.33, 95% CI 2-sided [0.09 to 0.56], Standard Error of Mean 0.121
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.1101, Mixed Models Analysis; LS mean difference = 0.23, 95% CI 2-sided [-0.05 to 0.52], Standard Error of Mean 0.146
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.0147, Mixed Models Analysis; LS mean difference = 0.32, 95% CI 2-sided [0.06 to 0.58], Standard Error of Mean 0.130
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.2032, Mixed Models Analysis; LS mean difference = 0.21, 95% CI 2-sided [-0.11 to 0.53], Standard Error of Mean 0.162
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.9345, Mixed Models Analysis; LS mean difference = -0.01, 95% CI 2-sided [-0.34 to 0.32], Standard Error of Mean 0.168
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.5968, Mixed Models Analysis; LS mean difference = -0.10, 95% CI 2-sided [-0.47 to 0.27], Standard Error of Mean 0.187
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 8]; Test type: Superiority; p = 0.7047, Mixed Models Analysis; LS mean difference = 0.06, 95% CI 2-sided [-0.26 to 0.39], Standard Error of Mean 0.166
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.8070, Mixed Models Analysis; LS mean difference = 0.04, 95% CI 2-sided [-0.27 to 0.35], Standard Error of Mean 0.157

39. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions 3 Levels (EQ-5D-3L) Score at Weeks 16 and 48
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions. Participants rated 5 aspects of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The mean of the summed score ranged from 1 to 3 with "1" corresponding to no problems and "3" corresponding to severe problems in the 5 dimensions, where higher score indicates more severe problems.
Time Frame: Baseline, Weeks 16 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 129 | 131
Units on a scale
  Week 16: Mobility | -0.23 (0.044) | -0.06 (0.044)
  Week 16: Self-Care | -0.21 (0.043) | -0.20 (0.043)
  Week 16: Usual Activities | -0.18 (0.046) | -0.09 (0.046)
  Week 16: Pain/Discomfort | -0.30 (0.036) | -0.12 (0.036)
  Week 16: Anxiety/Depression | -0.11 (0.048) | -0.10 (0.048)
  Week 48: Mobility | -0.32 (0.051) | -0.26 (0.050)
  Week 48: Self-Care | -0.33 (0.048) | -0.33 (0.047)
  Week 48: Usual Activities | -0.32 (0.053) | -0.34 (0.053)
  Week 48: Pain/Discomfort | -0.37 (0.047) | -0.36 (0.047)
  Week 48: Anxiety/Depression | -0.17 (0.054) | -0.21 (0.053)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Mobility: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.0030, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.28 to -0.06], Standard Error of Mean 0.055
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Self-Care: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.8970, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.055
Statistical Analysis 3: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Usual Activities: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.1437, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.20 to 0.03], Standard Error of Mean 0.058
Statistical Analysis 4: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Pain/Discomfort: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -0.18, 95% CI 2-sided [-0.27 to -0.09], Standard Error of Mean 0.046
Statistical Analysis 5: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16, Anxiety/Depression: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p = 0.8445, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.13 to 0.11], Standard Error of Mean 0.061
Statistical Analysis 6: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Mobility: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.3473, Mixed Models Analysis; LS mean difference = -0.06, 95% CI 2-sided [-0.19 to 0.07], Standard Error of Mean 0.064
Statistical Analysis 7: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Self-Care: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.9834, Mixed Models Analysis; LS mean difference = 0.00, 95% CI 2-sided [-0.12 to 0.12], Standard Error of Mean 0.059
Statistical Analysis 8: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Usual Activities: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.7364, Mixed Models Analysis; LS mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15], Standard Error of Mean 0.066
Statistical Analysis 9: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Pain/Discomfort: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.8075, Mixed Models Analysis; LS mean difference = -0.01, 95% CI 2-sided [-0.13 to 0.10], Standard Error of Mean 0.059
Statistical Analysis 10: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 48, Anxiety/Depression: Analysis performed using MMRM which included fixed effect of treatment group, visit, and treatment-group by visit interaction, stratification factor derived from clinical database, stratification-factor by visit interaction, baseline value, and baseline-value by visit interaction; Test type: Superiority; p = 0.5461, Mixed Models Analysis; LS mean difference = 0.04, 95% CI 2-sided [-0.09 to 0.17], Standard Error of Mean 0.067

40. Secondary Outcome: Change From Baseline in EuroQol Visual Analogue Scale (EQ-VAS) Score (mm) at Weeks 16 and 48
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions. Its second part included EQ-VAS. EQ-VAS recorded the participant's self-rated health on a VAS ranging from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state), with higher scores indicating better health state.
Time Frame: Baseline, Weeks 16 and 48
Population: FAS: included all participants who were randomized to the study and received at least one dose of the randomized investigational product (i.e., tofacitinib or placebo). Here, on-drug data was used and missing response was not imputed. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Here, "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 129 | 130
Millimeter (mm)
  Week 16: number analyzed (Participants) | 128 | 130
  Week 16 | 13.00 (1.840) | 2.89 (1.840)
  Week 48 | 20.64 (1.879) | 18.00 (1.862)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; Week 16: Analysis performed using ANCOVA model which included fixed effects of treatment group, stratification factor derived from clinical database, and baseline value; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 10.11, 95% CI 2-sided [5.52 to 14.70], Standard Error of Mean 2.331
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.2608, Mixed Models Analysis; LS mean difference = 2.63, 95% CI 2-sided [-1.97 to 7.24], Standard Error of Mean 2.337

41. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed Due to Health Problem at Weeks 16 and 48
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which Ankylosing Spondylitis affected work productivity and regular activities over the past 7 days. The questions are as follows: Q1 = currently employed; Q2 = hours missed due to health problems; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); Q6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent work time missed due to health problem was a subscale and calculated as: Q2/(Q2+Q4) for those who were currently employed. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Weeks 16 and 48
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 77 | 85
Units on a scale
  Week 16: number analyzed (Participants) | 74 | 81
  Week 16 | -3.65 (2.659) | 0.88 (2.622)
  Week 48 | -8.10 (2.136) | -5.79 (2.047)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p = 0.1784, ANCOVA; LS mean difference = -4.53, 95% CI 2-sided [-11.15 to 2.09], Standard Error of Mean 3.350
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.3651, Mixed Models Analysis; LS mean difference = -2.31, 95% CI 2-sided [-7.34 to 2.72], Standard Error of Mean 2.540

42. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Impairment While Working Due to Health Problem at Weeks 16 and 48
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which Ankylosing Spondylitis affected work productivity and regular activities over the past 7 days. The questions are as follows: Q1 = currently employed; Q2 = hours missed due to health problems; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); Q6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent Impairment while Working due to Health Problem was a subscale and calculated as: Q5/10 for those who were currently employed and actually worked in the past 7 days. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Weeks 16 and 48
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 75 | 82
Units on a scale
  Week 16: number analyzed (Participants) | 71 | 77
  Week 16 | -19.83 (2.274) | -6.94 (2.303)
  Week 48 | -25.35 (2.769) | -23.00 (2.656)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -12.89, 95% CI 2-sided [-18.59 to -7.19], Standard Error of Mean 2.884
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.4788, Mixed Models Analysis; LS mean difference = -2.36, 95% CI 2-sided [-8.92 to 4.21], Standard Error of Mean 3.318

43. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Overall Work Impairment Due to Health Problem at Weeks 16 and 48
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which Ankylosing Spondylitis affected work productivity and regular activities over the past 7 days. The questions are as follows: Q1 = currently employed; Q2 = hours missed due to health problems; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); Q6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent overall work impairment due to health problem was a subscale and calculated as: Q2/(Q2+Q4)+[(1- Q2/(Q2+Q4))×(Q5/10)] for those who were currently employed. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment.
Time Frame: Baseline, Weeks 16 and 48
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 75 | 82
Units on a scale
  Week 16: number analyzed (Participants) | 71 | 76
  Week 16 | -21.49 (2.508) | -7.64 (2.559)
  Week 48 | -27.63 (3.005) | -23.22 (2.890)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -13.85, 95% CI 2-sided [-20.18 to -7.52], Standard Error of Mean 3.202
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.2244, Mixed Models Analysis; LS mean difference = -4.41, 95% CI 2-sided [-11.56 to 2.74], Standard Error of Mean 3.613

44. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Activity Impairment Due to Health Problem at Weeks 16 and 48
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which Ankylosing Spondylitis affected work productivity and regular activities over the past 7 days. The questions are as follows: Q1 = currently employed; Q2 = hours missed due to health problems; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); Q6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent activity impairment due to health problem was a subscale and calculated as: Q6/10 for all respondents. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment.
Time Frame: Baseline, Weeks 16 and 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib | Placebo Then Tofacitinib
Number analyzed (Participants) | 129 | 131
Units on a scale
  Week 16 | -19.03 (1.969) | -5.63 (1.968)
  Week 48 | -27.37 (2.339) | -19.77 (2.310)
Statistical Analysis 1: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -13.40, 95% CI 2-sided [-18.30 to -8.50], Standard Error of Mean 2.488
Statistical Analysis 2: Comparison: Tofacitinib vs Placebo Then Tofacitinib; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0095, Mixed Models Analysis; LS mean difference = -7.60, 95% CI 2-sided [-13.32 to -1.88], Standard Error of Mean 2.905

ADVERSE EVENTS:
Time Frame: For the first 2 arms: (tofacitinib and Placebo [up to Week 16]): Baseline to Week 16 and for the next 2 arms (tofacitinib and placebo then tofacitinib [Day 1 to Week 48]): Baseline to Week 48
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who were randomized and received at least one dose of the investigational product (i.e., tofacitinib or placebo).
Groups:
- Tofacitinib: Up to Week 16: Participants received tofacitinib 5 mg tablets twice daily for 16 weeks.
- Placebo: Up to Week 16: Participants received tofacitinib matching placebo tablets, twice daily for 16 weeks.
- Tofacitinib: Day 1 to Week 48: Participants received tofacitinib 5 mg tablets twice daily for 48 weeks.
- Placebo Then Tofacitinib: Day 1 to Week 48: Participants received tofacitinib matching placebo tablets, twice daily for 16 weeks followed by tofacitinib tablets 5 mg, twice daily for next 32 weeks (i.e. up to Week 48).
Arm/Group | Tofacitinib: Up to Week 16 | Placebo: Up to Week 16 | Tofacitinib: Day 1 to Week 48 | Placebo Then Tofacitinib: Day 1 to Week 48
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/136 | 0/133 | 0/136
Serious Adverse Events (participants affected / at risk) | 2/133 | 1/136 | 7/133 | 2/136
Other Adverse Events (participants affected / at risk) | 23/133 | 26/136 | 51/133 | 52/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib: Up to Week 16 (N=133) | Placebo: Up to Week 16 (N=136) | Tofacitinib: Day 1 to Week 48 (N=133) | Placebo Then Tofacitinib: Day 1 to Week 48 (N=136)
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Condition aggravated (General disorders) | 0 | 1 | 0 | 1
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib: Up to Week 16 (N=133) | Placebo: Up to Week 16 (N=136) | Tofacitinib: Day 1 to Week 48 (N=133) | Placebo Then Tofacitinib: Day 1 to Week 48 (N=136)
Upper respiratory tract infection (Infections and infestations) | 14 | 10 | 21 | 18
Nasopharyngitis (Infections and infestations) | 9 | 10 | 11 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 2 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 10 | 8
Alanine aminotransferase increased (Investigations) | 0 | 0 | 8 | 2
Headache (Nervous system disorders) | 0 | 0 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 7
Protein urine present (Investigations) | 0 | 0 | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03502616/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03502616/SAP_001.pdf